## ASSESSMENT OF BIRTH OUTCOMES IN ESWATINI AFTER TRANSITION TO DOLUTEGRAVIR-BASED TREATMENT

## **Principal Investigators:**

Caspian Chouraya, MD, MSc; Michelle Gill, PhD, MPH; Bonisile Nhlabatsi, MPH

## **Institutions:**

Ministry of Health, Mbabane, Eswatini; Elizabeth Glaser Pediatric AIDS Foundation (EGPAF), Mbabane, Eswatini and Washington, DC, USA; George Washington University, Washington, DC, USA

Protocol Version 3.0, dated 26 August 2022

## Study Team

| Name, Surname and Contact Details | Roles and Responsibilities |
|---|---|
| Co-Principal Investigators | |
| Dr. Caspian Chouraya | Responsible for the in-country implementation |
| Country Director | of the evaluation, including staff recruitment, |
| EGPAF Eswatini | monitoring study progress, ensuring adherence |
| MVA Fund Office Park | to the scientific goal and ethical standards and |
| Mbabane, Eswatini | facilitating bidirectional communication with |
| Email: <a href="mailto:cchouraya@pedaids.org">cchouraya@pedaids.org</a> | evaluation team; ensuring transparent and |
| Phone: +268 24041811 | responsible program and financial management |
| | of the evaluation and overseeing data |
| | collection, analysis, report writing, and |
| | dissemination. Contributes to protocol |
| | development, overall conduct and management |
| | and the scientific integrity of the study at |
| | country level. Ensures government and |
| | stakeholder involvement and coordination. |
| Dr. Michelle Gill | Responsible for protocol development, overall |
| Associate Research Director | conduct (including ethical), management, and |
| EGPAF US | the scientific integrity of the study at global |
| 1140 Connecticut Ave NW, Suite 200 | level. Monitors study progress to ensure study |
| Washington, DC 20036 USA | objectives will be met. Leads interpretation of |
| Email: mgill@pedaids.org | study findings, manuscript writing and |
| Phone: +1 2024488403 | dissemination and results utilization. Liaises |
| | with in-country PI and other investigators and |
| | the donor. |
| MOH Principal | Investigator |
| Bonisile Nhlabatsi | Contributes to the implementation of the study, |
| Program Manager | guiding protocol development and study |
| Ministry of Health, Eswatini | implementation to ensure alignment with |
| Sexual Reproductive Health Unit (SRHU) | national policies and priorities and ensure |
| Email: thandazabn@yahoo.com | transparent bidirectional communication with |
| Phone: +268 76114263/ +268 24050003 | relevant units within the MOH at regional and |
| | national levels. |
| Co-Invest | igators |
| Dr. Lynne Mofenson | Provides support to the study team, both global |
| Senior HIV Technical Advisor | and in-country. Will provide technical |
| EGPAF US | leadership in the implementation of research |
| Email: <u>lmofenson@pedaids.org</u> | and evaluation projects, and contribute to |
| Phone: +1 2024077970 | results interpretation and write-up, development |
| | of publications, and results utilization. |

| Dr. Vincent Tukei | Advises on clinical study issues and |
|---|---|
| Research Director | interpretation of clinical data. Liaises with |
| EGPAF Eswatini | EGPAF and MOH on program and study |
| Email: vtukei@pedaids.org | related issues. Will help to ensure that |
| Phone: +268 78086511 | experiences from the study are used to inform |
| 1 Hone. 1200 70000311 | the ongoing national surveillance system and |
| | government and stakeholder involvement and |
| | coordination. |
| Philisiwe Khumalo | Contributes to the day-to-day implementation |
| Senior Public Health Evaluation Manager | of study activities, including translation of |
| EGPAF Eswatini | evaluation tools and SOPs, training and |
| Email: pkhumalo@pedaids.org | supervision, ethics and regulatory compliance, |
| Phone: +268 24048081 | management of data abstraction/collection |
| 1 Hone. 1200 24040001 | activities, quality, and analysis and |
| | dissemination and serve as the liaison for |
| | communication and coordination with ethical |
| | review boards at the Ministry of Health. |
| Dr. Heather Hoffman | Responsible for developing statistical analysis |
| The George Washington University | plan, lead analysis of data, and contribute to the |
| Milken Institute School of Public Health | write up of study findings. |
| Biostatistics and Bioinformatics Department | write up or study findings. |
| Email: hhoffman@gwu.edu | |
| Phone: +1 2029948587 | |
| MOH Co-inv | estigators |
| | esugutors |
| Ntombikayise Dlamini-Madlopha | Contribute to the design and implementation of |
| Maternal and Newborn Officer | the study, guide protocol development and |
| Ministry of Health, Eswatini | study implementation to ensure alignment with |
| Sexual Reproductive Health Unit (SRHU) | national policies and priorities and ensure |
| Emial: <u>kayisedee@gmail.com</u> | transparent bidirectional communication at |
| Phone: +268 76086890 | health facility level. Also contribute to the |
| | overall management of data |
| | abstraction/collection activities, data quality, |
| | and analysis and dissemination activities. |
| Wiseman Mngometulu | Contribute to the design and implementation of |
| PMTCT Focal, Community Mentor Mother | the study, guide the development and |
| Coordinator | implementation to ensure alignment with |
| Ministry of Health, Eswatini | national policies and priorities and ensure |
| Sexual Reproductive Health Unit (SRHU) | transparent bidirectional communication at |
| Email: wisdomwisey2@gmail.com | health facility level. Also contribute to data |
| Phone: +268 76187748 | quality assurance, review and interpretation |
| | and dissemination activities. |
| Nompumelelo Mthunzi | Contribute to the design and implementation of |
| Senior Monitoring and Evaluation Analyst | the study, guide the development and |

Ministry of Health, Eswatini

Strategic Information Department (SID)

Email: <a href="mpumiemthunzi@gmail.com">mpumiemthunzi@gmail.com</a>
Phone: +268 24047252, +268 76210119

implementation to ensure alignment with national policies and priorities and ensure transparent bidirectional communication at health facility level. Also contribute to data quality assurance, review and interpretation and dissemination activities.

## Table of Contents

| Acronyms | 6 |
|-----------------------------------|----|
| Protocol Summary | 7 |
| Background & Scientific Rationale | 9 |
| Study Objectives | 12 |
| Study Design & Methods | 12 |
| Study Design Summary | 12 |
| Site Selection | 13 |
| Study Population | 14 |
| Sample Size Calculation | 14 |
| Study Procedures | 15 |
| Enrolment: | 15 |
| Chart abstraction: | 16 |
| Interviews with women | 17 |
| Training | 18 |
| Study Variables and Definitions | 19 |
| Data Management | 21 |
| Confidentiality Protections | 22 |
| Statistical Analysis Plan | 23 |
| Ethical Considerations | 24 |
| Informed Consent Procedures | 24 |
| Risks and Benefits | 25 |
| Request for Consent Waiver | 25 |
| Serious Adverse Events Reporting | 26 |
| Compensation for Participation | 26 |
| Ethical Review | 26 |
| Limitations | 26 |
| Dissemination and Utilization | 26 |
| Estimated Study Timeline | 27 |
| References | 28 |

## Acronyms

ANC Antenatal care

APMR ART Patient Monitoring and Reporting
APR Antiretroviral Pregnancy Registry

ART Antiretroviral therapy

ARV Antiretroviral

CMIS Client management information system

DTG Dolutegravir EFV Efavirenz

EGPAF Elizabeth Glaser Pediatric AIDS Foundation

EHHRRB Eswatini Health and Human Research Review Board

IPD Inpatient Department
IRB Institutional Review Board
LMP Last menstrual period
MOH Ministry of Health

NNRTI Non-nucleoside reverse-transcriptase inhibitor

NRTI Nucleoside reverse transcriptase

NTD Neural tube defect OPD Outpatient Department PI Protease inhibitor

PIN Personal identity number

PMTCT Prevention of Mother-to-Child Transmission

PrEP Pre-exposure prophylaxis

SID Strategic Information Department SRHU Sexual Reproductive Health Unit

WHO World Health Organization

## **Protocol Summary**

Dolutegravir (DTG) is a second-generation integrase inhibitor that has demonstrated improved virologic efficacy and tolerance compared to efavirenz (EFV)-based first-line ART. Initial data in May 2018 from the Tsepamo study in Botswana had suggested a potential ~9-fold increase in risk of neural tube defects (NTD) among infants delivered to women receiving DTG at the time they became pregnant. However, in the most recent analysis through March 2022, NTD prevalence had stabilized at a low level, 0.11% (10 NTD in 9,460 exposures to DTG at conception); this is now the same as the NTD prevalence of 0.11% with non-DTG ART at conception (25 NTD in /23,664 births) and is compared to 0.07% in women without HIV infection (108 NTD in 170,723 births). Based on previous data from this study in 2020, demonstrating an earlier decrease in NTD prevalence, and updated risk-benefit analyses demonstrating that the benefits of DTG significantly outweigh the potential risks, the World Health Organization recommends DTG as a preferred first-line drug for treatment, but also indicates continued surveillance is needed to more definitively confirm or refute the NTD signal among women of reproductive potential.

To contribute to the evidence base on birth defects among women on DTG at conception and to support the national birth surveillance system that can be used to determine the rate of birth defects in the general population and evaluate outcomes of emergent therapies, we will be conducting an observational study at five high volume hospitals in Eswatini, in which birth defect and other data will be collected at the time of delivery for all women. The overall aim of this study is to evaluate the birth outcomes of HIV-positive women who are receiving DTG or other ARV drug regimens. The primary research objectives are to: 1) determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-positive women on DTG at conception; 2) determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-negative women; and 3) determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-positive women on non-DTG ART at conception.

Data collection over an approximate 24-month period will involve two main components. The first is birth surveillance designed to capture the deliveries of all women presenting to study hospitals, including HIV-positive women with DTG exposure both before and during pregnancy or on another or no ART regimen and HIV-negative women as well as any stillbirths. Mothers' pregnancy history, birth outcomes, and HIV and ART information (as applicable) will be collected from existing clinic registers, reporting forms and databases. Secondly, more detailed information on health history, risk factors, and descriptions of birth defects and classification by clinical staff, will be collected through interviews and photographs with consenting mothers whose children have been identified by clinical staff to have major external birth defects at the time of delivery, or in the event of a medical abortion following the identification of a serious fetal birth defect

through ultrasonography. This information will be sent to an external pediatric specialist for a final confirmatory diagnosis.

NTD will be the primary study outcome. Key secondary outcome variables include other major and surface birth defects and other pregnancy outcomes that could be associated with ARV exposure, such as preterm delivery, low birthweight and stillbirths. The primary analysis will be descriptive, to determine the proportion of NTD among infants delivered by HIV-positive women on DTG at conception and HIV-negative women. Exploratory statistical investigations may be performed for birth defects or other outcomes among women living with HIV receiving DTG at conception, women living with HIV receiving non-DTG ART at conception, and women without HIV infection. If assumptions are met for NTD prevalence and the expected number of deliveries, one year of surveillance from these hospitals could provide the sample size needed to rule-out a relatively rare event like an NTD: approximately 10,000 women on DTG at conception.

Results will be disseminated by EGPAF to the Eswatini MOH at regional and national levels and other key stakeholders in-country as well as to a global audience to share information critical to our understanding of birth defects and other birth outcomes, among women on DTG at conception and in the general population.

## Background & Scientific Rationale

Ensuring people living with HIV are on optimal ART regimens is a critical component to reaching the UNAIDS 95-95-95 goals by 2030 [1]. Dolutegravir (DTG) is a second-generation integrase inhibitor that has demonstrated improved virologic efficacy and tolerance compared to efavirenz (EFV)-based first-line ART [2, 3]. DTG has a high barrier to resistance, and in the face of growing transmitted and acquired drug resistance, especially to non-nucleoside reverse-transcriptase inhibitors (NNRTIs) like EFV, DTG offers strong first-line therapy [4, 5]. DTG has also been shown to be effective and safe when used for second-line therapy in combination with an optimized nucleoside reverse transcriptase (NRTI) backbone in individuals with virologic failure on NNRTI or protease inhibitor (PI)-based first-line regimens [6-8]. Two randomized clinical trials in pregnant women starting ART after the first trimester have demonstrated that DTG ART more rapidly decreased viral load than EFV ART, with a significantly larger proportion of women having undetectable viral load at delivery with DTG than EFV ART [9, 10].

However, in May 2018, investigators from the Tsepamo study, a multi-site surveillance of birth outcomes for HIV-positive and HIV-negative women at hospitals in Botswana reported a potential signal for neural tube defects (NTD) with use of DTG ART at conception [11]. Four NTD were identified in 426 (0.94%) women receiving DTG at the time they became pregnant. This was significantly greater than all other comparison groups, including women on non-DTG ART regimens at the time of conception, 14 NTD/11,300 deliveries, prevalence 0.12%; starting DTG during pregnancy, 0 NTD/2,812 deliveries; and HIV-negative women, 61 NTD/66,057 deliveries, prevalence 0.09%. The study expanded from eight to 18 sites, covering 72% of all births in Botswana. Repeat analysis of data through March 2019 demonstrated a decrease in NTD prevalence with receipt of DTG at conception to 0.30% (five NTD among 1,683 deliveries) [12]. While the prevalence of NTD declined from the initial report, the NTD prevalence remained significantly higher than observed with non-DTG ART at conception (0.10%), EFV at conception (0.04%), or DTG started during pregnancy (0.04%), or in HIV-uninfected women (0.08%). Additionally, the Botswana Ministry of Health and Wellness expanded surveillance of birth outcomes at 22 selected non-Tsepamo health facilities, expanding coverage to 92% of all births in Botswana when combined with Tsepamo sites [13]. From October 2018 through March 2019, at the MOH sites, one NTD was identified among 152 women receiving DTG at conception (prevalence 0.66%) compared to no NTD among 381 HIV-positive women receiving non-DTG ART at conception and two among 2,328 HIV-uninfected women (0.09%).

A more recent analysis of the Tsepamo study including data through April 2020 was presented at the International AIDS Conference in July 2020. The prevalence of NTD with DTG at conception further decreased to 0.19% (seven NTD/3,591 deliveries), remaining stable at this rate from September 2019 through April 2020 [14]. In comparison, NTD prevalence with non-DTG ART

at conception was 0.11% (21 NTD/19,361 deliveries), with the prevalence difference between DTG vs non-DTG at conception no longer statistically significantly different (prevalence difference 0.09%, 95% CI -0.03, 0.30%). The prevalence difference with DTG at conception did remain significantly higher than EFV at conception (eight NTD/10,958 deliveries, 0.07%, prevalence difference 0.12%), DTG started during pregnancy (two NTD/4,581 deliveries, 0.04%, prevalence difference 0.15%), and HIV-uninfected women (87 NTD/119,630 deliveries, 0.07%, prevalence difference 0.12%). Finally, the most recent results from the Tsepamo study, including data through March 2022 was presented at the International AIDS Conference in July 2022. NTD prevalence had stabilized at a low level, 0.11% (10 NTD in 9,460 exposures to DTG at conception); this is now the same as the NTD prevalence of 0.11% with non-DTG ART at conception (25 NTD in /23,664 births) and is compared to 0.07% in women without HIV infection (108 NTD in 170,723 births). The prevalence of NTD in infants born to women on DTG at conception does not substantially differ from other exposure groups; prevalence difference between DTG versus non-DTG at conception (0.00%, 95% CI -0.07, 0.10) and versus HIV-uninfected women (0.04%, 95% CI -0.01, 0.13).

Outside of the Botswana studies, one other NTD has been reported in the January 2020 Antiretroviral Pregnancy Registry (APR) out of 382 women receiving DTG at the time of conception (prevalence 0.26%) [15]. However, most reports in the APR come from higher income countries, most with national food folate fortification, which has been shown to be associated with a decline in population prevalence of NTD [16, 17]. In Brazil, a retrospective chart review of all women with pregnancies and possible DTG exposure included in the national antiretroviral therapy database was conducted; the results found no NTDs during the study period in women conceiving on either DTG (n=382) or EFV (n=1,045) as a comparator [18]. However, two NTD were reported post-hoc in women conceiving on DTG, bringing the estimated NTD prevalence with DTG at conception to 0.18% [18, 19]. Brazil has national food folate fortification, and this NTD prevalence with DTG at conception is higher than the population NTD prevalence estimate of 0.06% [20].

Thus, the available data suggest that if DTG at conception is associated with an increased risk of NTD, this risk is likely a ~2 to 3-fold increase over the overall population rates, and not the ~9-fold increase suggested by the initial Tsepamo data in May 2018. To provide perspective on the prevalence increase observed with non-genetic factors associated with an increased risk of NTD, maternal diabetes is associated with a 2 to 10-fold increase in NTD, maternal obesity a 1.5 to 3.5-fold increase, maternal hyperthermia a 2-fold increase, low maternal red blood cell folate levels a 4-fold increase, and receipt of valproate around the time of conception a 10-fold increase [21, 22].

<sup>&</sup>lt;sup>1</sup>Zash R et al. Update on neural tube defects with antiretroviral exposure in the Tsepamo study, Botswana. 24th International AIDS Conference, Montreal, abstract PELBB02, 2022.

Based on the decreased NTD prevalence in the updated Tsepamo study and updated risk-benefit analyses demonstrating that the benefits of DTG significantly outweigh the potential risks [5, 23, 24], the World Health Organization (WHO) recommends DTG as a preferred first-line drug for treatment as well as a preferred second-line drug in combination with an optimized NRTI backbone in individuals failing NNRTI or protease inhibitor –based therapy [25]. The 2019 guidelines note that women should be provided with information about benefits and risks to make an informed choice regarding the use of DTG or other ART, and that continued surveillance is needed to more definitively confirm or refute the NTD signal.

Eswatini is an optimal context in which to conduct birth surveillance and generate additional data in sub-Saharan Africa in a country without folate food fortification. The adult HIV prevalence is one of the highest in the world at 27% and is 35% among pregnant women [26, 27]. The facility delivery rate is 87.7% [28]. This relatively small country has 12 public hospitals, allowing for focused efforts in facility-level capacity building and data system strengthening in a subset of high volume hospitals to allow for robust data collection of birth outcomes in the country. Eswatini began transition of HIV-positive adolescents and adults, including women of reproductive potential, to DTG-based first- and second-line ART in April 2019. DTG introduction was gradual, particularly among women in this group, in an effort to first use existing EFV stock. However, transition is expected to ramp up in 2021 and thus, preconception DTG exposures will occur during the next couple years in Eswatini, making it an ideal country to institute further birth outcome surveillance to provide additional reliable data from Africa to refute or confirm the existing NTD association.

EGPAF has been supporting the Kingdom of Eswatini since 2003 to prevent mother-to-child HIV transmission (PMTCT) and to provide HIV and AIDS care and treatment services to HIV-positive children and adults. Currently, EGPAF supports 65 health facilities in Hhohho and Shiselweni regions of Eswatini with PMTCT, HIV prevention (voluntary medical male circumcision, pre-exposure prophylaxis [PrEP]), HIV testing and counseling, ART and tuberculosis services. Together with the Ministry of Health (MOH) and other implementing partners, EGPAF has been leading efforts to strengthen birth outcomes monitoring, which will help ensure this surveillance study is well integrated into national health programming.

With planned broad transition of programs to DTG-based ART for first- and second-line treatment, it will be important to have in place sentinel surveillance to evaluate birth outcomes in women who become pregnant while receiving DTG or any new drug regimen. Through this effort, EGPAF will enhance the existing surveillance program through sentinel surveillance conducted as part of the study in five high-volume public hospitals. The system will allow for the collection of data on preconception DTG exposures and birth defects by capturing deliveries from all HIV-positive and HIV-negative women, primarily using existing facility sources. This surveillance will strengthen and improve upon efforts by the Eswatini MOH to introduce national routine pregnancy outcome and infant monitoring, helping to ensure the sustainability of such a system to evaluate new drugs

and interventions as they come to market, such as long-acting antiretrovirals for HIV treatment and prevention. Furthermore, there are currently no population-based estimates of birth defects in Eswatini. In addition to its utility in providing the comparative group for evaluating the effects of DTG exposure, these data will be useful for the country as a whole in describing the general burden of birth defects.

## **Study Objectives**

The overall aim of this study is to evaluate the birth outcomes of HIV-positive women who are receiving DTG or other ARV drug regimens. The following primary research objectives will be addressed in selected hospitals in Eswatini:

- 1. To determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-positive women on DTG at conception.
- 2. To determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-negative women.
- 3. To determine the proportion of neural tube defects among live and stillborn infants delivered by HIV-positive women on non-DTG ART at conception.

The secondary research objectives are described below.

- 1. To determine the general prevalence of major external birth defects among all live and stillborn infants regardless of maternal HIV or ART status.
- 2. To describe pregnancy outcomes (e.g., all major and surface birth defects, preterm delivery, low birthweight, miscarriages) among women by HIV status, by ART regimen, by timing of exposure to DTG (pre- or post-conception), and other factors such as maternal age at delivery and gravida.

## Study Design & Methods

### Study Design Summary

This is an observational study at sentinel sites to evaluate the birth outcomes of women receiving the standard of care for ART treatment and the outcomes of HIV-negative women, with data collected at one time point for all women, at the time of delivery. Collecting data on all women who deliver at these sentinel sites with detailed information on any newborns with identifiable

birth defects will be critical to our understanding of birth outcomes and any birth defects. This will be achieved by conducting birth outcomes surveillance, with data collection planned on all deliveries during an approximate 24-month period. The target population includes all HIV-positive women with DTG exposure both before and during pregnancy, HIV-positive women on another or no ART regimen, and HIV-negative women delivering at selected hospitals. Detailed information will be collected through chart abstraction for all women, and through interviews and photographs with consenting mothers whose children have been identified to have major external birth defects

NTD will be the primary study outcome. Key secondary outcome variables include other major and surface birth defects and other pregnancy outcomes that could be associated with ARV exposure, such as preterm delivery, low birthweight and stillbirths. The primary analysis will be descriptive, to determine the proportion of NTD among infants delivered by HIV-positive women on DTG at conception, HIV-negative women, and any available women not on DTG. Exploratory statistical investigations and modeling may be performed for birth defects or other outcomes among the groups described in secondary objective #2 provided there are sufficient sub-group numbers to do so. This will also depend on the extent of DTG transition at the time of data collection, particularly for comparisons of HIV-positive women on non-DTG regimens and those initiating DTG during pregnancy.

## Site Selection

The study will be conducted in high-volume public hospitals (Table 1) across all four regions of Eswatini. Five out of the 12 hospitals in the country with the highest number of deliveries in 2020 were selected purposively. In January 2020 to December 2020, there were 20,501 deliveries in the selected hospitals and 6,393 deliveries among HIV-positive women who were on ART in antenatal care (ANC) [29]. Of the HIV-positive women on ART in ANC, 85% were on ART at the first visit, resulting in an estimated 5,434 women on ART at the time of conception in these five hospitals for the one-year period [26]. Assuming uptake of DTG will range from 65% to 90% for the women enrolled during the study period and that the delivery numbers for HIV positive women will be similar to previous programmatic numbers, this is estimated to yield 3,145 deliveries of women on DTG at conception. If assumptions are met or exceeded for NTD prevalence and the expected number of deliveries after one year of surveillance from these hospitals, approximately two years of enrollment could provide the sample size needed to rule-out a relatively rare event like an NTD (see Table 2).

Table 1. Study hospitals and number of deliveries, January to December 2020

| No | Region | Hospital | # of | # of HIV | # of HIV | Estimated # of |
|----|--------|----------|------------|----------|----------|----------------|
| | | | deliveries | positive | positive | women on |
| | | | | women | women | DTG at |
| | | | | | on ART | conception* |

| 1 | Hhohho | Mbabane Government<br>Hospital | 5,579 | 1,768 | 1,767 | 872 |
|---|---|---|---|---|---|---|
| 2 | Manzini | Raleigh Fitkin Memorial Hospital | 5,534 | 1,979 | 1,978 | 961 |
| 3 | Manzini | Mankayane Government Hospital | 2,516 | 7,14 | 712 | 378 |
| 4 | Lubombo | Good Shepherd<br>Hospital | 3,659 | 1,104 | 1,097 | 531 |
| 5 | Shiselweni | Hlathikhulu Hospital | 3213 | 828 | 825 | 403 |
| | Total | | 20,501 | 6,393 | 6,379 | 3,145 |

<sup>\*</sup>Based on assumptions and previous programmatic estimates

### Study Population

For capture of routine pregnancy information, the study population is defined as all women delivering infants at selected hospitals in Eswatini, including women delivering stillborn infants and those who would have miscarriages or medical abortions due to identified congenital defects. A subset of this population will be recruited for additional data collection. Inclusion criteria for this subset are: (1) a birth defect as identified by a midwife or other clinician at the study hospital and (2) willing to provide informed consent. For the additional data collection component, women of any age will be considered eligible. Adolescents less than 18 years of age, defined as emancipated minors due to their pregnancy/motherhood status, will be asked to provide informed consent for themselves.

## Sample Size Calculation

The sample size target will be based on updated Tsepamo study findings from 2022, which found an NTD prevalence of 0.11% (10/9,460 deliveries) compared to earlier data from 2019 which found a prevalence of 0.30% (5/1,683 deliveries) among women receiving DTG ART at conception [12]. When the sample size is between 7,500-10,000 for the exposure group of interest, a two-sided Wilson score-based 95% confidence interval for a single proportion will have a precision of 0.00083-0.00098 for an expected NTD prevalence of 0.11% among deliveries to women with DTG at conception exposure with a probability of at least 95% (Table 2)[30]. Sample sizes based on the prevalence for the other two groups using the latest Tsepamo study findings are also presented (0.07% for HIV-negative women and 0.11% for HIV-positive women not on DTG). As we expect the enrollment number for HIV-negative women to be higher than the other groups and the number of HIV-positive women on non-DTG regimens at conception to be low as DTG transition efforts mature, precision estimates are presented according to these expectations. Larger sample sizes will increase the power and decrease the type I error in the statistical models used to address secondary objective 2; therefore, we will enroll everyone during the study period. Sample sizes are provided in the table below based on varying proportions and precision.

Table 2. Sample sizes based on assumed proportions (0.0007, 0.0011) and precision ranges

| Proportion | Precision (Half-Width) | Sample Size (N) | Probability |
|---------------|------------------------|-----------------|-------------|
| HIV-negative | 0.0013 | 3800 | 0.946 |
| | 0.0014 | 3600 | 0.957 |
| 0.0007 | 0.0015 | 3400 | 0.966 |
| | 0.0016 | 3200 | 0.973 |
| HIV-positive | 0.00083 | 10000 | 0.968 |
| on DTG at | 0.00085 | 9500 | 0.962 |
| conception | 0.00087 | 9000 | 0.955 |
| | 0.00090 | 8500 | 0.946 |
| 0.0011 | 0.00095 | 8000 | 0.965 |
| | 0.00098 | 7500 | 0.958 |
| HIV-positive | 0.0029 | 1500 | 0.974 |
| on non-DTG | 0.0032 | 1400 | 0.980 |
| at conception | 0.0034 | 1300 | 0.985 |
| | 0.0035 | 1200 | 0.955 |
| 0.0011 | 0.0036 | 1100 | 0.965 |

As there is some uncertainty with respect to the number of deliveries that will be observed among women receiving DTG ART at conception, enrollment numbers will be reviewed monthly for progress towards the study sample size to assess the likely trajectory for achieving the target sample size. All deliveries will be captured to help ensure we are positioned to detect an association between DTG preconception exposure and NTD, if one exists, and to be able to describe the prevalence of NTD in the general population.

## Study Procedures

### Enrolment:

Data collection will involve two main components: 1) birth surveillance designed to capture the deliveries of all women presenting to the five study hospitals and 2) interviews with women and photographs taken of their newborns with possible defects identified at birth. For each delivery, midwives or data collectors will complete a paper-based version of the study enrollment log (or master linking document) by writing in the date of admission, date of delivery, unique patient identifiers (e.g., Personal Identity Number [PIN], ANC and ART as applicable), ANC health facility name and the woman's name and her phone number, which are necessary to locate and link women's information in the registers and other sources (e.g., CMIS, APMR) and confirm her contact information in the case of duplicated/multiple records. To ensure that delivery data are captured in real-time (including weekends and overnight), facility-based nurse midwives will assist at the first point of data collection, particularly during off-work hours, when feasible. Per routine practice, nurse midwives will examine the infant for external birth defects; examinations of stillborns will be conducted if feasible. For each woman's entry on the log, the outcome of this examination will be documented, to capture whether or not a major external birth defect was identified. A generic term (e.g., 'determination') and an accompanying numeric response code will be used so those outside the study would not know the meaning of the code, to avoid capturing

any sensitive information in this log. This would then help to determine the next data collection step for each woman: recruit, consent, and interview to capture more detailed information on her health history and risk factors if there is a birth defect; if not, the data clerk will proceed with data abstraction. Additional procedures for each of these two steps are described below.

#### Chart abstraction:

Trained data collectors will be stationed at each study hospital and will be primarily responsible for data collection of still- and live-born deliveries at maternity, and any miscarriages or medical abortions due to identified congenital defects of women presenting to the facilities (Gynecology/outpatient department [OPD]/inpatient department [IPD]) to the extent possible. Each day, data collectors will review the enrollment logs completed by midwives and cross-reference those forms with the clinic registers to verify that all deliveries have been captured. They will abstract basic information about the mother, child, pregnancy and delivery using registers, patient handheld cards, and other paper-based or electronic sources, such as the national client management information system (CMIS) and the ART Patient Monitoring and Reporting (APMR), to the extent necessary, and enter into a study record using an electronic form loaded onto an electronic device. Since routine information will be collected from the existing records, and does not include any primary data collection with participants, the activity presents no more than minimal risk of harm to participants and a waiver of consent is requested.

The main study data sources used in hospitals will be the maternity and perinatal registers and the ANC card. Data, which are not available in the hospital registers or the ANC card, will be accessed in the following way:

• Data from women's electronic database entries will be extracted and integrated into their study records. This will be done by data collectors at hospitals using the onsite databases or by study staff accessing them offsite (e.g., at the EGPAF national office). For the latter, this is likely to occur when additional data collection support is needed or when the older version of an electronic database like CMIS, APMR, or the health management information system (HMIS) needs to be accessed, for example, when women received care at an ART clinic that has not yet been updated to the current electronic data capture system. Variables include PrEP regimen and start and stop dates for women who were HIV negative at the time and for women with HIV, ARV drugs taken at current regimen (as applicable) and date of last menstrual period (LMP) for women presenting to the gynecological ward or other department with miscarriages or for recommended medical abortions and for women presenting to maternity if it has not already been captured by midwives.

As part of completion of the enrollment log for women presenting to maternity, midwives or data collectors will capture the women's LMP from her handheld ANC card (if she has brought her card and this information is documented in her card), as this is critical to determining primary

outcomes, and other information as needed (see Table 3). Receipt of PrEP in pregnancy will also be captured on the log, and a 'yes' response will prompt data collectors or the larger study team to extract regimen and start and stop dates from electronic sources as needed and as described above for the women's study record.

Information about miscarriages (or spontaneous abortions, defined as < 28 weeks gestation), will also be captured to the extent possible, but will be dependent on women's self-report and presentation to the gynecological ward. Similarly, information about medically induced abortions will also be collected as feasible (described further below). Data collectors will make regular, frequent visits to the ward or other departments co-located at the same hospital as the maternity to check for any miscarriages (which may be found in the gynecological inpatient and outpatient registers or improvised registers) or medical abortions. Clinic staff may also notify study team members of women potentially meeting study criteria outside of the maternity ward. Similar information will be abstracted for women with miscarriages and abortions (to the extent it is available) and live or still births.

#### Interviews with women

A woman who delivers an infant with an identified major external birth defect will be referred by clinic staff and recruited for enrollment into a separate study component. Because women who have abortions will only be recruited for the study if the pregnancy was terminated due to the presence of a birth defect detected by imaging, attempts will also be made to interview them. If this is not feasible, for instance if the woman has already been discharged or the midwife is unavailable, her information will be abstracted from existing records, similar to the procedure for miscarriages as described above, plus information on the identified congenital defect. These data may be collected retrospectively (while still within the study period) or prospectively.

If she is willing to hear more about the study, she will undergo an informed consent process. Nurses and data collectors will be trained in the administration of informed consent, and either may perform this task. Women will be interviewed for more in-depth information on her HIV testing and ART history, other medical history of selected conditions (e.g., diabetes, malaria, TB) and potential teratogenic exposures. Data will be verified from the women's handheld patient cards and other medical records as available. Accompanying photographs of the infant will also be taken (with consent) from multiple perspectives to provide a complete picture of the defect.

As routine practice, doctors based at the maternities should examine any infant identified by the nurse midwife as having an external defect and consult on the diagnosis. As part of surveillance, existing EGPAF mentors and the study team will support efforts to standardize and strengthen this practice. The interview responses, which will include relevant details of the major structural abnormality through closed and open-ended questions, and photographs (if available), will be sent to an external expert/specialist, for a final confirmatory diagnosis by the study coordinator or other study team member. This expert will have training in medical genetics or a similar field and have

experience with these types of reviews for other studies or registries. The specialist will review the information (first stripped of HIV and ART status) and diagnosis made by the site level clinical team. It will not include the woman's name, contact information or the hospital name; she will be identified by her study identification number only. Healthcare workers will receive feedback on the diagnoses made by the specialist. If the diagnosis by the specialist differs from the diagnosis made by the clinical staff, healthcare workers in study sites may contact the mother (with permission and phone number obtained at the time of the interview) to inform her of the final diagnosis and provide any further information or referrals as needed and appropriate.

Below is a figure that summarizes the flow of information for possible birth defects identified at surveillance sites, including reporting to the donor (ViiV Healthcare) and to the institutional review boards (IRBs).

Figure 1. Flow Chart for Possible Major External Birth Defects Identified at Surveillance Site



#### **Training**

As part of the study, health providers (doctors, nurses) in each hospital maternity will receive training to further strengthen their skills in examination and identification of birth defects. The study coordinator will also provide support to midwives at maternities for surveillance activities. The study coordinator and investigators will conduct regular monitoring visits to the hospitals to provide mentorship on performing examinations to ensure birth defects are accurately classified

and to review surveillance forms against facility records for quality assurance. In addition, mentorship and supportive supervision are already provided by implementing partners (including EGPAF) and by the MOH on a regular basis. Training and ongoing supportive supervision will be provided to nurse midwives and other providers at study hospitals to strengthen documentation practices, in addition to skills building for conducting examinations and identifying birth defects.

## Study Variables and Definitions

For all deliveries/births, routine data will be captured on mother's pregnancy history, birth outcomes, and HIV and ART information as applicable. Variables to be collected will include:

- Mother's age, gravidity, parity, LMP, and HIV status
- Pregnancy outcomes: stillbirth (≥ 20 weeks), prematurity (< 37 weeks), delivery mode, infant birth weight, any major surface birth defects, including NTD, and neonatal death before discharge
- If HIV-positive: ART regimen at time of conception (ARVs, date initiated) and any changes through delivery (ARVs, start/stop dates).
- If HIV-negative: receipt of PrEP in pregnancy (start/stop dates), PrEP regimen

Table 3 below presents the variables to be collected through surveillance on all women and probable variable sources. They are subject to change, and will be ultimately determined by what is routinely collected under the program, as we are relying on existing data. Tool versions and instructions for completion may change over time and we will align our data collection accordingly.

Table 3. Illustrative variables to be collected for routine surveillance (all women), by likely source

| Variables | | Source(s) |
|---|---|---|
| Pregnancy and | Mother's age | Maternity register, Perinatal register |
| HIV history | ANC facility | Maternity register, ANC card |
| | Last menstrual period | ANC card |
| | Gravidity | Maternity register |
| | Parity | Maternity register, Perinatal register |
| | HIV status and date of last test prior | Maternity register, Perinatal register |
| | to L&D | |
| | HIV retesting (eligibility, testing date | Maternity register |
| | and result) | |
| | HIV testing if not tested previously | Maternity register |
| | (testing date and result) | |
| | Gestational age at first ANC | Perinatal register |
| Birth outcomes | Gestational age at delivery | Perinatal register |
| | Mode of delivery | Maternity register, Perinatal register |
| | Date of delivery | Maternity register, Perinatal register |
| | Stillbirth (FSB, MSB) | Maternity register, Perinatal register |
| | Sex of baby | Maternity register, Perinatal register |

| | Weight at birth | Maternity register, Perinatal register |
|---|---|---|
| | Single or multiple birth | Free form text in maternity register* |
| | Neonatal death before discharge: | Perinatal register |
| | cause, baby age at death | - |
| ART/PrEP | Current ART regimen and date | CMIS, APMR, Perinatal register, handheld |
| | started | ART card |
| | ART regimen at time of conception | CMIS, APMR, handheld ART card |
| | (if different from above), start/stop | |
| | dates | |
| | Any other ART regimen taken during | CMIS, AMR, handheld ART card |
| | pregnancy (if applicable), start/stop | |
| | dates | |
| | Receipt of PrEP in pregnancy | ANC card |
| | Current PrEP use, regimen, start/stop | CMIS, ANC card, APMR |
| | dates | |
| | | ges and medically induced abortions** |
| Pregnancy and | Mother's age | Gyn OPD/IPD registers, ANC card |
| HIV history | Last menstrual period | CMIS, ANC card |
| | Gravidity | Gyn/OPD/IPD registers, ANC card |
| | Parity | Gyn/OPD/IPD registers, ANC card |
| | Pregnancy condition | Gyn/OPD/IPD registers, ANC card |
| | HIV status | Gyn/OPD/IPD registers, ANC card, CMIS, |
| | | APMR, handheld ART card |
| ART/PrEP | On ART | Gyn/OPD/IPD registers, ANC card, CMIS, |
| | | APMR, handheld ART card |
| | Current ART regimen and date | CMIS, APMR, ANC card, handheld ART |
| | started | card |
| | ART regimen at time of conception | CMIS, APMR, ANC card, handheld ART |
| | (if different from above), start/stop | card |
| | dates | |
| | Any other ART regimen taken during | CMIS, APMR, ANC card, handheld ART |
| | pregnancy (if applicable), start/stop | card |
| | dates | |
| | Current PrEP use, regimen start/stop | CMIS, APMR, ANC card |
| 7:110 | dates | |
| Birth defect | Birth defect and description | Ultrasound scan report |
| (abortions only) | | |

<sup>\*</sup>Will capture to the extent that this is appropriately documented.

For the primary analysis, outcomes will be defined as follows:

**HIV-positive status:** women with a documented positive result in the perinatal and/or maternity register or other clinical source record.

**HIV-negative status**: women with the last HIV test result recorded during pregnancy or labor and delivery as negative.

<sup>\*\*</sup>Abortions due to identified congenital defects will only be captured under surveillance if it is not possible to conduct an interview

**DTG at conception:** (for women on DTG-based regimens): determined using the date of initiation of DTG and date of LMP or gestational age at delivery (if LMP not available). Given the uncertainty around LMP and dates of conception, we are defining ART at conception as maternal ART that started up to 8 weeks after the calculated LMP date, which would be up to 6 weeks after the estimated date of conception. This will help to ensure we include the first 4 weeks of gestation, the defined period for neural tube closure.

**NTD**: definite (confirmed by photograph) or probable (diagnosed on the basis of a description but with no photograph) myelomeningocele, meningocele, encephalocele, anencephaly with or without craniorachischisis or iniencephaly.

Other birth defects: Using the parameters defined by the Tsepamo study, other abnormalities identified by routine surface examination before hospital discharge will be classified as major external structural malformations if they are deemed to be significant from a clinical, surgical or cosmetic standpoint [12]. Also as in Tsepamo, surface examinations will not include those of the inside of the mouth, auscultation of the heart, or testing for inguinal hernias, undescended testes, or hip dysplasia. Other diagnostics, such as imaging, may be used to make a birth defect determination for women who ultimately undergo a medically induced abortion as a result of a birth defect identified in utero. Ultrasounds are occasionally used at study hospitals at the request of patients or under certain circumstances, though chromosomal testing, mutation analysis and autopsy data will not be used.

## Data Management

Data will be entered directly into ODK-X database (from tablet or any other configured electronic devices) using existing paper-based and electronic clinical record sources. Data collectors will be primarily responsible for birth surveillance while data collectors and nurse midwives will be responsible for interviews with women and taking photographs. Both will work together to help ensure every woman meeting study eligibility criteria is captured. Everyone responsible for collecting data or supervising collection will be trained on protocol specific procedures, research ethics and data entry procedures into ODK-X. Branching and skip patterns as well as logic checks and reasonable ranges will be built into data collection tools to help assure data quality. In addition, data collected for the study may need to be triangulated using multiple clinic sources, patient handheld cards, and electronic databases for relevant variables; the study team may request providers help to reconcile inconsistencies across sources.

Experienced EGPAF data management staff will oversee data entry and maintain the study database. The database will be stored on a secure web-based server using the ODK-X platform,

which has built-in encryption capabilities. All electronic devices used in the study will be password protected and access to the ODK-X application will include another level of authentication.

Data will be synchronized with the secure cloud-based server maintained by EGPAF Global, ideally on a daily basis or later (e.g., weekly) when internet connectivity is intermittent. For data that may need to be extracted from electronic sources at the EGPAF Mbabane office, the data manager or other data staff will be able to update entries to the most up-to-date database and make other modifications as needed. The study database will be automatically backed up daily on OneDrive-based repository. The backups will synchronize automatically at multiple specified times during the day. In case of data loss in the primary database in country, these backups will be used for data recovery. The in-country data manager will be responsible for the daily operations of the database, including verifying that the data are synchronizing properly between point of data collection and the database. The global data manager will support the in-country team in terms of building additional validation controls as needed, verifying that the backups are synchronizing properly on the server and routine maintenance of the server. Access to the EGPAF server will be restricted to authorized study personnel.

### **Confidentiality Protections**

There is a minimal risk of confidentiality breach. Clinic and other ID numbers, names and contact numbers will be collected to ensure our ability to link data for a complete study record and carry out quality assurance practices. In addition, by virtue of their presence in the clinic and data abstraction activities from existing clinic records, data collectors and other study team members as part of study monitoring, will view individual health information. However, identifying information will not be contained in the same dataset with study-related information from the abstraction and interviews; this information will only be identified by a unique study identification (ID) number.

At each hospital, the study team will maintain a master enrollment log that permits linking of the participant through their ID numbers, name and contact number used for health services delivery, to their unique study number. As described above, data collectors and midwives will be responsible for completing the log. Unique study ID numbers will be preprinted on the enrollment logs. This master log will be kept in a locked cabinet in a locked office with limited access at study sites. Data collectors will also enter selected information (PIN, clinic numbers, names, phone numbers, and study ID numbers) into an abbreviated electronic version of the log loaded onto the electronic device. Only selected members of the study team will have access to the paper and electronic master documents based on the need to facilitate data collection. The electronic version will have even greater restricted access and will be used primarily for quality assurance and to enter any updates to the records that can only be done through accessing national databases from a central (office) location; data collectors will only view/access the electronic log for their respective sites. In addition, all study team members will sign a data handling and confidentiality agreement and complete an online ethics course certification. Data will also be stored in password-protected

systems or devices, with prompts to change passwords on a regular basis. Finally, to the extent possible, data abstraction will occur in a private location of the health facility to minimize any risk of unauthorized viewing of medical records.

Separate enrollment logs will be maintained for women who participate in interviews and will include participant names, the unique study ID number assigned to them and the date consented and enrolled into the study. If they agree, the log will also include their phone number to be contacted in case additional follow-up information is deemed necessary to provide after the specialist's review. Participant names and contact information will not be on any study documents linked to their interview responses nor in the study database. To minimize the risk of someone inadvertently hearing women's responses, the study team will work with hospital managers to identify private areas for interviews, such as a separate consultation room.

The enrollment logs will be destroyed after completion of data analysis. Other paper-based study documents, namely the signed consent forms for women participating in interviews, will be retained for five years after completion of the study. After that time, the documents will be destroyed and the in-country PI or designee will document the destruction.

Information provided to the specialist on birth defects will be stripped of any identifiers and shared securely with appropriate safeguards in place (e.g., password-protection, secure link instead of email). They will have access to this information until the final study analyses are completed, then we will request the specialist to document the destruction/deletion of all related study materials.

## Statistical Analysis Plan

Summary statistics will be calculated for all variables of interest to describe the sample. Specifically, means and standard deviations or medians and interquartile ranges (depending on the distribution of the data) as well as minima and maxima will be calculated for all continuous variables. Frequency counts and percentages will be reported for all categorical variables.

Primary Objectives 1, 2, and 3: The proportion of NTD among all live and stillborn infants delivered by (1) HIV-positive women on DTG at conception and (2) HIV-negative women will be calculated as the number of births with NTD divided by the total number of births for each group of women, and (3) HIV-positive women on non-DTG ART at conception. The 95% confidence intervals around these proportions will be calculated with the Wilson Score method, which is appropriate for small proportions close to zero. The difference in the proportions between the three groups will be estimated along with the corresponding 95% confidence interval based on the Newcombe method. These analyses will be conducted both with and without NTD identified through ultrasound for women who underwent medically induced abortions. Statistical inference will only be made if there is sufficient power to do so.

**Secondary Objective 1:** The general prevalence (proportion) of major external birth defects among all live and still born infants regardless of maternal HIV or ART status will be calculated as the number of births with major external birth defects divided by the total number of births to all women. The 95% confidence intervals around the prevalence of these birth defects will be calculated with the Wilson Score method.

Secondary Objective 2: Frequencies and proportions of pregnancy outcomes (e.g., all major and surface birth defects, preterm delivery, low birthweight) will be calculated along with 95% Wilson Score confidence intervals for subgroups of women based on HIV status, ART regimen, timing of exposure to DTG (pre- or post-conception), and timing of exposure to any other ART regimen. Estimates of differences in proportions among HIV-positive women will be considered as follows: (1) Women who started on DTG ART preconception and those who started on non-DTG regimen preconception; (2) women who started on DTG preconception and those who started on DTG during pregnancy; and (3) women who started on DTG preconception and those who started a non-DTG regimen during pregnancy. Finally, all HIV-positive women on any ART regimen will be compared to HIV-negative women. Differences in these proportions between the subgroups of women will be examined with simple (unadjusted) and multiple (adjusted) logistic regression or log-binomial models. Relative risk (risk ratios) will be reported along with their corresponding 95% confidence intervals. If reliable statistical estimates cannot be generated, due to a small number of cases, we will use Firth's penalized maximum likelihood approach. Adjusted models will control for factors such as maternal age at delivery and gravida. All potential covariates will be pre-defined in a separate data analysis plan.

## **Ethical Considerations**

#### Informed Consent Procedures

Written informed consent will be obtained by midwives or study staff trained in consenting procedures prior to the collection of any primary study data. Before conducting an interview, they will explain the study to the participant using the informed consent form in their preferred language (siSwati or English). This will include the purpose of the study, the risks and benefits of participation and how risks will be mitigated. They will explain that participation is voluntary and it is their choice to participate in the study; participants will be assured that they may refuse to participate or refuse to answer any questions and it will not affect their receipt of any health services. The consent form will be read clearly to participants; literate participants or witnesses of illiterate participants will be asked to read along. Participants will have the opportunity to ask any questions regarding study procedures. Once the consent form has been read and the participant feels all their questions and/or concerns have been addressed, literate participants will be asked to sign and date the consent form in the appropriate signature block. For those who are illiterate, a

thumbprint will be used to indicate consent and a witness will observe the consent process, sign and date the form to certify that the participant has been read the consent on that day and voluntarily agreed to take part in the study. Participants will be offered a copy of the informed consent form, which includes study team's contact numbers, in case they have any additional questions about participation.

Women with deliveries who consent for the study will be asked if they agree to 1) participate in an interview, 2) have photographs taken of her child (children for multiple births) to help classify the birth defect, and 3) be followed up later if the specialist reviewing her case has a different diagnosis than the maternity or other pertinent information to share. However, women may still participate in the study if they only agree to #1 or #2; if they agree to one or both of these components, they may also still participate in the study, even if they do not consent to #3.

#### Risks and Benefits

This observational study has minimal risk, with the primary risk being a breach of confidentiality. Ways to address this and the risk of privacy breaches have been described above in a previous section. Secondly, women participating in interviews could also feel uncomfortable or upset by the questions on their previous health history, use of drugs or other therapies, or their HIV status, particularly as they are being questioned after learning of a major birth defect in their child or undergoing an abortion. The midwives and other study staff who may be involved in this study component will be trained in non-biased interview techniques and undergo role-playing in training sessions to hone this practice. Participants will also be assured that they do not have to answer any question that they do not feel comfortable responding to, and that they may leave the study at any time.

There will be no direct benefits to participants from taking part in this study. However, the information provided by participants will add make a valuable contribution to the international and national evidence base on birth defects and risk factors, which could help to improve pregnancy and birth outcomes in the future for other women and their children.

#### Request for Consent Waiver

Other than the primary data collected from women with probable or definite birth defects, surveillance data will be available through routine collection of clinical data during the provision of medical care. No additional information will be collected outside of what is routinely recorded in patient records during standard medical care. For this component, there will be no direct interaction with the patients by the data collectors or other study team members for the purposes of the study. Therefore, a waiver of informed consent is being requested for the following reasons according to the U.S. Code of Federal Regulations (CFR 46.116(f)):

- 1. The research presents no more than minimal risk of harm to subjects,
- 2. The waiver or alteration will not adversely affect the rights and welfare of the subjects; and

3. The research could not practicably be carried out without the waiver or alteration (given the number of deliveries to captured as necessitated by this study design).

## Serious Adverse Events Reporting

While they are not anticipated, any serious adverse event related to the study, and which the study team is made aware of, will be reported promptly to the IRBs and the donor in accordance with their respective procedures. Reporting of any birth defects and stillbirths among women on DTG will be reported to the donor per Figure 1 above. This information will be summarized in annual reports to the IRBs. Any suspected or confirmed breaches in confidentiality will also be reported to the IRBs and the study facility will be notified as appropriate.

## Compensation for Participation

Study participants will not be paid to participate in the study, nor will they be provided with incentives.

#### **Ethical Review**

This protocol will be reviewed by the Eswatini Health and Human Research Review Board (EHHRRB) and an IRB in the US.

## Limitations

As this study relies heavily on routinely collected data, the primary study limitation is possible incomplete recording by health providers and inaccuracies in the records. As described above, the study team will support nurse midwives and other providers at study hospitals to strengthen documentation practices to mitigate this risk. Study staff will perform routine quality assurance checks and resolve missing and inaccurate data entries to the extent possible through ongoing data cleaning and frequent site monitoring. Secondly, as this study takes place at hospitals only, we will not be able to capture the outcomes of home deliveries. However, the facility delivery rate in the country is about 88%. Similarly, women who experience miscarriages may not present to the clinic, so we will likely underrepresent this number. Finally, during the interviews with women, there may be a certain degree of social desirability or recall biases as they try to remember for instance the name and timing of a particular medication they took, especially after they have just learned of a birth defect in their newborn or fetus. Interviewers will be trained to employ tools such as calendars, reminders of memorable events like holidays and use photographs or descriptions of certain drugs to help stimulate one's memory. They will also be trained to ask questions and receive responses in a way that does not imply judgement.

## Dissemination and Utilization

The Eswatini MOH will work closely with EGPAF to disseminate results at regional and national levels and other key stakeholders in-country through study-specific meetings and via existing platforms, such as technical working group and research advisory committee meetings. The MOH will be involved throughout the study preparation and implementation stages, through MOH investigators (from the Sexual Reproductive Health Unit), Health Research and Innovations Unit, and Epidemiology and Disease Control Unit to help ensure that data serve the country's needs for birth surveillance and that results can inform the birth surveillance network for Eswatini going forward. At regional and global levels, findings from this study will be shared across other EGPAF programs and with the donor. Abstract(s) will be submitted for consideration at national and international meetings and manuscript(s) will be submitted to an international peer-reviewed journal.

The results will inform the ongoing national surveillance program, through the provision of feedback on the quality and completeness of key indicators that could be considered for any national tool refinements and the surveillance process itself (e.g., data collection, clinic flow, etc.). As relevant, data on DTG-based ART and other regimens will also be shared with the Eswatini National AIDS Program to contribute to future discussions on national ART guideline updates for women of child-bearing age.

## **Estimated Study Timeline**

Below is an estimated study timeline, starting from the time of receipt of IRB approval. Once approval of the protocol package has been obtained from Eswatini and US IRBs, the study duration is estimated to be 30 months, with approximately one month to develop standard operating procedures, train midwives and other study staff and prepare facilities, 24 months for data collection and approximately five months following data collection to clean, analyze and disseminate the final data. Interim data analysis, writing and dissemination activities will also be conducted while data collection is ongoing.

| | | QUARTER (Q) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ACTIVITY | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 |
| Study training and site preparation | X | | | | | | | | | |
| Data collection | X | X | X | X | X | X | X | X | X | |
| Data cleaning and analysis | | | | | X | | | | X | |
| Write-up of findings | | | | | X | X | | | X | X |
| Dissemination | | | | | | X | | | | X |

## References

- 1. UNAIDS. On the fast-track to an AIDS free generation. Geneva: UNAIDS; 2016 [cited 2018 April 21]. Available from: <a href="www.unaids.org/sites/default/files/media\_asset/GlobalPlan2016\_en.pdf">www.unaids.org/sites/default/files/media\_asset/GlobalPlan2016\_en.pdf</a>.
- 2. Walmsley S, Baumgarten A, Berenguer J, Felizarta F, Florence E, Khuong-Josses MA, et al. Brief Report: Dolutegravir Plus Abacavir/Lamivudine for the Treatment of HIV-1 Infection in Antiretroviral Therapy-Naive Patients: Week 96 and Week 144 Results From the SINGLE Randomized Clinical Trial. J Acquir Immune Defic Syndr. 2015;70(5):515-9.
- 3. Venter WDF, Sokhela S, Simmons B, Moorhouse M, Fairlie L, Mashabane N, et al. Dolutegravir with emtricitabine and tenofovir alafenamide or tenofovir disoproxil fumarate versus efavirenz, emtricitabine, and tenofovir disoproxil fumarate for initial treatment of HIV-1 infection (ADVANCE): week 96 results from a randomised, phase 3, non-inferiority trial. The lancet HIV. 2020;7(10):e666-e76.
- 4. Vitoria M, Hill A, Ford N, Doherty M, Clayden P, Venter F, et al. The transition to dolutegravir and other new antiretrovirals in low-income and middle-income countries: what are the issues? Aids. 2018;32(12):1551-61.
- 5. Phillips AN, Bansi-Matharu L, Venter F, Havlir D, Pozniak A, Kuritzkes DR, et al. Updated assessment of risks and benefits of dolutegravir versus efavirenz in new antiretroviral treatment initiators in sub-Saharan Africa: modelling to inform treatment guidelines. The lancet HIV. 2020;7(3):e193-e200.
- 6. Hamers RL. Dolutegravir for second-line antiretroviral therapy. The Lancet Infectious diseases. 2019;19(3):218-9.
- 7. Aboud M, Kaplan R, Lombaard J, Zhang F, Hidalgo JA, Mamedova E, et al. Dolutegravir versus ritonavir-boosted lopinavir both with dual nucleoside reverse transcriptase inhibitor therapy in adults with HIV-1 infection in whom first-line therapy has failed (DAWNING): an open-label, non-inferiority, phase 3b trial. The Lancet Infectious diseases. 2019;19(3):253-64.
- 8. Waitt C, Orrell C, Walimbwa S, Singh Y, Kintu K, Simmons B, et al. Safety and pharmacokinetics of dolutegravir in pregnant mothers with HIV infection and their neonates: A randomised trial (DolPHIN-1 study). PLoS medicine. 2019;16(9):e1002895.
- 9. Kintu K, Malaba TR, Nakibuka J, Papamichael C, Colbers A, Byrne K, et al. Dolutegravir versus efavirenz in women starting HIV therapy in late pregnancy (DolPHIN-2): an open-label, randomised controlled trial. The lancet HIV. 2020;7(5):e332-e9.
- 10. Chinula L, Brummel SS, Ziemba L, Stranix-Chibanda L, Coletti A, Krotje C, et al. Safety and efficacy of DTG vs EFV and TDF vs TAF in pregnancy: IMPAACT 2010 trial. Conference on Retroviruses and Opportunistic Infections; Boston, Mass. 2020.
- 11. Zash R, Makhema J, Shapiro RL. Neural-Tube Defects with Dolutegravir Treatment from the Time of Conception. The New England journal of medicine. 2018;379(10):979-81.
- 12. Zash R, Holmes L, Diseko M, Jacobson DL, Brummel S, Mayondi G, et al. Neural-Tube Defects and Antiretroviral Treatment Regimens in Botswana. The New England journal of medicine. 2019;381(9):827-40.
- 13. Raesima MM, Ogbuabo CM, Thomas V, Forhan SE, Gokatweng G, Dintwa E, et al. Dolutegravir Use at Conception Additional Surveillance Data from Botswana. The New England journal of medicine. 2019;381(9):885-7.
- 14. Zash R, Holmes L, Diseko M, Jacobson D, Mayondi G, Isaacson A, et al. Update on neural tube defects with antiretroviral exposure in the Tsepamo study, Botswana. 23rd International AIDS Conference Virtual, 2020.

- 15. Antiretroviral Pregnancy Registry Steering Committee. Antiretroviral Pregnancy Registry Interim Report for 1 January 1989 through 31 January 2020 Wilmington, NC: Registry Coordinating Center; 2020. Available from: www.APRegistry.com].
- 16. Amarin ZO, Obeidat AZ. Effect of folic acid fortification on the incidence of neural tube defects. Paediatric and perinatal epidemiology. 2010;24(4):349-51.
- 17. De Wals P, Tairou F, Van Allen MI, Uh SH, Lowry RB, Sibbald B, et al. Reduction in neural-tube defects after folic acid fortification in Canada. The New England journal of medicine. 2007;357(2):135-42.
- 18. Pereira GFM, Kim A, Jalil EM, Fernandes Fonseca F, Shepherd BE, Veloso VG, et al. Dolutegravir and pregnancy outcomes in women on antiretroviral therapy in Brazil: a retrospective national cohort study. The lancet HIV. 2021;8(1):e33-e41.
- 19. Abrams E, Myer L. Lessons from dolutegravir and neural tube defects. The lancet HIV. 2021;8(1):e3-e4.
- 20. Santos LM, Lecca RC, Cortez-Escalante JJ, Sanchez MN, Rodrigues HG. Prevention of neural tube defects by the fortification of flour with folic acid: a population-based retrospective study in Brazil. Bulletin of the World Health Organization. 2016;94(1):22-9.
- 21. Avagliano L, Massa V, George TM, Qureshy S, Bulfamante GP, Finnell RH. Overview on neural tube defects: From development to physical characteristics. Birth defects research. 2019;111(19):1455-67.
- 22. Crider KS, Devine O, Hao L, Dowling NF, Li S, Molloy AM, et al. Population red blood cell folate concentrations for prevention of neural tube defects: Bayesian model. BMJ (Clinical research ed). 2014;349:g4554.
- 23. Dugdale CM, Ciaranello AL, Bekker LG, Stern ME, Myer L, Wood R, et al. Risks and Benefits of Dolutegravir- and Efavirenz-Based Strategies for South African Women With HIV of Child-Bearing Potential: A Modeling Study. Annals of internal medicine. 2019;170(9):614-25.
- 24. Estill J, Bertisch B. More evidence for dolutegravir as first-line ART for all. The lancet HIV. 2020;7(3):e154-e5.
- 25. World Health Organization. Update of recommendations on first- and second-line antiretroviral regimens. Geneva, Switzerland: World Health Organization; 2019. Available from: <a href="https://apps.who.int/iris/bitstream/handle/10665/325892/WHO-CDS-HIV-19.15-eng.pdf?ua=1">https://apps.who.int/iris/bitstream/handle/10665/325892/WHO-CDS-HIV-19.15-eng.pdf?ua=1</a>].
- 26. Eswatini Ministry of Health. Swaziland Health Information Management System 2. 2017.
- 27. Eswatini Ministry of Health. Annual HIV Programs Report. 2018.
- 28. Central Statistical Office and UNICEF. Multiple Indicator Cluster Survey (MICS) Final Report 2014. Mbabane, Eswatini: Central Statistical Office and UNICEF; 2016. Available from: <a href="https://mics-surveys-surveys-">https://mics-surveys-</a>
- prod.s3.amazonaws.com/MICS5/Eastern%20and%20Southern%20Africa/Eswatini/2014/Final/Swaziland%202014%20MICS%20Final%20Report English.pdf].
- 29. EGPAF. Programmatic data. 2020.
- 30. Watts DH. Teratogenicity risk of antiretroviral therapy in pregnancy. Current HIV/AIDS reports. 2007;4(3):135-40.

Eswatini Birth Outcomes Study

# Assessment of Birth Outcomes in Eswatini after Transition to Dolutegravir-Based Treatment Chart Abstraction Form for live births, stillbirths and miscarriages

| M | ATERNITY NAME | | | |
|---|---|---|---|---|
| | | | MBABANE ( | GOVERNMENT HOSPITAL 1 |
| | | | RALEIGH FITKI | N MEMORIAL HOSPITAL 2 |
| | | | Goo | OD SHEPHERD HOSPITAL 3 |
| | | | | HLATIKHULU HOSPITAL 4 |
| | | | Mankayane ( | GOVERNMENT HOSPITAL 5 |
| DA | ATA COLLECTOR'S NAME/ID: | | DAY / MONTH / YEAR OF ABSTRACTION | ON: |
| | , | | | |
| N/ | AME: | | // | 2 0 |
| | | <del></del> | | |
| ID | ): | | | |
| D/ | ATA COLLECTION POINT: | | | |
| | W. Collection Court | MATERNITY | | |
| | OPD | /GYNECOLOGY | | |
| # | Variables | Response Opti | | Directions |
| | Pregnan | cy and HIV his | story, Source: registers | |
| 1. | Date of admission | | | |
| | (dd/mm/yyyy) | | // | |
| 2. | Mother's age | | years 1 | |
| | 2 11: | Unk | nown/not documented 87 | |
| 3. | Gravidity | Links | # of pregnancies 1 nown/ not documented 87 | |
| 4. | Parity | Oliki | # of births 1 | |
| 4. | Parity | Unk | nown/not documented 87 | |
| 5. | Last menstrual period (LMP) | | | |
| 6. | Gestational age at L&D booking | | weeks, days 1 | |
| | | Don't | know/not documented 287 | |
| | Not applicable for miscarriages/ | | N/A 🗌 99 | |
| | medical induced abortions | | | |
| 7. | HIV status at L&D/admission | | HIV positive 1 | |
| | | | HIV negative 2 | |
| | | Limb | Never tested for HIV 4 | |

| 8. | Tested for HIV at L&D (indicate | Yes 1 | |
|---|---|---|---|
| | yes if there is a date of HIV test | No 🔲 2 | SKIP TO Q |
| | entered) | Unknown/not documented 87 | SKIP TO Q |
| | , | N/A ∐ 99 | SKIP TO Q |
| | Not applicable for miscarriages/ | | |
| | medically induced abortions | | |
| 9. | HIV test result at L&D | HIV positive 1 | |
| | | HIV negative 2 | |
| | Not applicable for miscarriages | Inconclusive 3 | |
| | Not applicable for miscarriages | N/A 99 | |
| 10. | Date of most recent HIV test prior | / 1 | |
| | to L&D | Unknown/not documented 🗌 87 | |
| | (dd/mm/yyyy) | N/A 🗌 99 | |
| | Not applicable for miscarriages | | |
| | Bir | rth outcomes, Source: registers | |
| 11. | Birth outcome | Live birth 1 | |
| | | Stillbirth 2 | |
| | | Miscarriage 3 | If miscarriage or |
| | | Medically induced abortion 4 | abortion, go to Q22 |
| 12. | Single or multiple birth | Single 1 | For options 2 and 3, |
| 12. | Single of multiple birth | Twin 2 | form will return to Q12 |
| | Not applicable for missarringes/ | Triplet 3 | to ask for each |
| | Not applicable for miscarriages/ | N/A ☐ 99 | |
| | medically induced abortions | N/A ☐ 99 | subsequent child while |
| | | | retaining the same |
| | | | maternal information |
| 13. | Gestational age at delivery | weeks, days 1 | |
| | | Unknown/not documented 87 | |
| 14. | Mode of delivery | Normal vaginal delivery (NVD) 🔲 1 | |
| | | Assisted vaginal delivery (AVD) 🗌 2 | |
| | | Elective C-section (ELCS) 3 | |
| | | Emergency C-section (EMCS) 4 | |
| 15. | Date of delivery | | |
| | (dd/mm/yyyy) | /1 | |
| 16. | If stillbirth | FSB (fresh) 1 | |
| | | MSB (macerated) 2 | |
| | | N/A – live birth 99 | |
| 17. | Sex of baby | Male 1 | |
| | 1 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | Female 2 | |
| | | Ambiguous 3 | |
| 18. | Weight at birth | grams | |
| 10. | weight at biltil | Unknown/not documented 87 | |
| 19. | Neonatal death before discharge | Yes 1 | |
| 19. | iveonatai deatii belole disclidige | No 2 | SKIP TO Q |
| 20 | Causes of infant death | | JAIF TO Q |
| 20. | Causes of illiant death | 1 | |

| 21. Infant age at death | Unknown/not documented 87 Q25 | | | Unknown/not documented 🗌 87 | |
|---|---|---|---|---|---|
| 22. If miscarriage or abortion, date of miscarriage/abortion (dd/mm/yyyy) | 22. If miscarriage or abortion, date of miscarriage/abortion (dd/mm/yyyy) Different from admission 1 Different from admission date: | 21. | Infant age at death | hours | For all responses go to |
| miscarriage/abortion (dd/mm/yyyy) 23. Gestational age at time of | miscarriage/abortion Different from admission date: (dd/mm/yyyy) | | | Unknown/not documented 🗌 87 | Q25 |
| Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. ART regimen Yes 1 No 2 SKIP to Q 2 | (dd/mm/yyyy) | 22. | If miscarriage or abortion, date of | Same as date of admission 1 | |
| Unknown/not documented | Unknown/not documented | | miscarriage/abortion | Different from admission date: | |
| 23. Gestational age at time of miscarriage/abortion | 23. Gestational age at time of miscarriage/abortion | | (dd/mm/yyyy) | // | |
| miscarriage/abortion 24. Pregnancy condition 25. Was a birth defect identified? 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). 27. ART regimen 28. First two drugs ('NRTI backbone') ABC/3TC 1 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 STIP It is to all infants | miscarriage/abortion 24. Pregnancy condition 25. Was a birth defect identified? 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., precalampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). 27. ART regimen 28. First two drugs ('NRTI backbone') ART yegimen: 29. Third drug listed in the CURRENT ART regimen: 29. Third drug listed in the CURRENT ART regimen: 20. Third drug listed in the CURRENT ART regimen: 20. Third drug listed in the CURRENT ART regimen: 20. Third drug listed in the CURRENT ART regimen: 20. Third drug listed in the CURRENT ART regimen: 21. ART regimen: 22. ART regimen: 23. ART regimen: 24. ART regimen: 25. ART regimen: 26. Comments: Please use this and in the current | | | Unknown/not documented 2 87 | |
| 24. Pregnancy condition 25. Was a birth defect identified? Ves | 24. Pregnancy condition 25. Was a birth defect identified? 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). 27. ART regimen 28. First two drugs ('NRTI backbone') SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 29. Third drug listed in the CURRENT ART regimen: 29. Third drug listed in the CURRENT ART regimen: 29. Third drug listed in the CURRENT ART regimen: 29. Third drug listed in the CURRENT ART regimen: 29. Third drug listed in the CURRENT ART regimen: 29. Third drug listed in the CURRENT SURRENT ART 29. Third drug listed in the CURRENT SURRENT 20. SURRENT SURRENT SURRENT 20. SURRENT SURRENT SURRENT 21. SURRENT SURRENT 22. SURRENT SURRENT SURRENT 23. SURRENT SURRENT 24. SURRENT SURRENT 25. SURRENT SURRENT 26. SURRENT SURRENT 27. SURRENT SURRENT 28. SURRENT SURRENT 29. SURRENT SURRENT SURRENT 20. SURRENT SURRENT 20. SURRENT SURRENT 21. SURRENT SURRENT 22. SURRENT | 23. | Gestational age at time of | # of births 1 | |
| 25. Was a birth defect identified? Ves | 25. Was a birth defect identified? Yes | | miscarriage/abortion | Unknown/not documented 🗌 87 | |
| 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 2 TDF/3TC 3 3 Other, specify: | Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. | 24. | Pregnancy condition | | |
| 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 2 TDF/3TC 3 3 Other, specify: | Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. | | | | |
| 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 2 TDF/3TC 3 3 Other, specify: | Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. | 25 | Was a hirth defect identified? | Ves 1 | |
| 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 No 2 SKIP to Q | 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes: Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 AZT/3TC 2 TDF/3TC 3 Isted in the CURRENT ART regimen: Other, specify: 88 Unknown/not documented 87 29. Third drug listed in the CURRENT RT regimen: EFV 2 ATV/r 3 LPV/r 4 DTG 5 DRV 6 Other, specify: 88 Unknown/not documented 87 | 25. | was a sirtif defect identified: | | |
| 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 TDF/3TC 3 Other, specify: | 26. Comments: Please use this section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen ART regimen Yes | | | Unknown/not documented 🔲 87 | |
| section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 | section to indicate any additional relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes | | | N/A 🗌 99 | |
| relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 2 TDF/3TC 3 3 TDF/3TC 3 3 TDF/3TC 3 3 TDF/3TC 3 88 | relevant information found in source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen ART regimen Yes | 26. | | | |
| source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: | source documents, including maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen ART regimen Yes | | - | | |
| maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). **Applies to all infants/birth outcomes.** **Antiretroviral Therapy (ART), Sources: registers, electronic database** 27. ART regimen | maternal complications (e.g., preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 TDF/3TC 3 TDF/3TC 3 TDF/3TC 3 TDF/3TC 3 NDF/3TC 3 | | | | |
| preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 listed in the CURRENT ART regimen: Other, specify: | preeclampsia, diabetes, etc.) or child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 TDF/3TC 3 Other, specify: 88 Unknown/not documented 87 29. Third drug listed in the CURRENT ART EFV 2 ATV/r 3 LPV/r 4 DTG 5 DRV 6 Other, specify: 88 Unknown/not documented 87 | | | | |
| child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 listed in the CURRENT ART AZT/3TC 2 regimen: Other, specify: | child's condition (e.g., birth defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Pes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 1 AZT/3TC 2 TDF/3TC 3 Other, specify: 88 Unknown/not documented 87 29. Third drug listed in the CURRENT ART EFV 2 ATV/r 3 LPV/r 4 DTG 5 DRV 6 Other, specify: 88 Unknown/not documented 87 | | | | |
| defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: | defect, jaundice, prematurity). Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen 28. First two drugs ('NRTI backbone') ABC/3TC 1 | | | | |
| Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') ABC/3TC 1 listed in the CURRENT ART | Applies to all infants/birth outcomes. Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen 28. First two drugs ('NRTI backbone') ABC/3TC | | | | |
| Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: | Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes | | defect, jaundice, prematurity). | | |
| Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: | Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes | | | | |
| Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: Other, specify: 1 AZT/3TC 2 TDF/3TC 3 Other, specify: 88 | Antiretroviral Therapy (ART), Sources: registers, electronic database 27. ART regimen Yes | | | | |
| 27. ART regimen Yes 1 No 2 SKIP to Q 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: Other, specify: 88 | 27. ART regimen | | | way (ART) Carrier was interestable all atmospic datab | |
| 28. First two drugs ('NRTI backbone') ABC/3TC ☐ 1 listed in the CURRENT ART regimen: AZT/3TC ☐ 2 Other, specify: B8 | No | 27 | | | ase<br>I |
| 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: ABC/3TC 1 AZT/3TC 2 TDF/3TC 3 Other, specify: 88 | 28. First two drugs ('NRTI backbone') listed in the CURRENT ART regimen: Other, specify: | 27. | AKT regimen | l <u> </u> | SKIP to O |
| listed in the CURRENT ART regimen: AZT/3TC 2 TDF/3TC 3 Other, specify: | listed in the CURRENT ART regimen: Other, specify: | 28. | First two drugs ('NRTI backbone') | | |
| Other, specify: 88 | Other, specify: | | = : | l <u>=</u> | |
| Other, specify: <u></u> 88 | Other, specify: | | regimen: | <u> </u> | |
| Unknown/not documented [_] 87 | 29. Third drug listed in the CURRENT ART regimen: ART regimen: | | S | l — | |
| | ART regimen: EFV | | | Unknown/not documented [_] 87 | |
| 29 Third drug listed in the CURRENT NVP 1 | ART regimen: EFV | 29 | Third drug listed in the CURRENT | NVP ☐ 1 | |
| | ATV/r 3 LPV/r 4 DTG 5 DRV 6 Other, specify: 88 Unknown/not documented 87 | 23. | _ | | |
| 7.11.1 regimen: | DTG | | , and regiment | l <u>=</u> | |
| LPV/r ☐ 4 | Other, specify: | | | LPV/r ☐ 4 | |
| | Other, specify: 88 Unknown/not documented 87 | | | | |
| | Unknown/not documented 87 | | | _ | |
| Inknown/not documented 07 | 130 1 Date started (TIRRENT ART 1 Known 1 1 1 | 30 | Date started CURRENT ART | | |
| | | 50. | | | |
| 30. Date started CURRENT ART Known 1 | regimen Date / / | | - regimen | | |
| 30. Date started CURRENT ART Known 1 1 regimen Date:// | | | | | |
| 30. Date started CURRENT ART Known 1 | regimen Date: / / | | - | | |
| 30. Date started CURRENT ART Known 1 | | | | Unknown/not documented 87 | |

| 31. | If unknown, when was current | During pregnancy 1 | |
|---|---|---|---|
| | regimen started? | Before pregnancy 2 | |
| | S | Unknown/not documented 🗌 87 | |
| 32. | Changes in ART regimen in the | Yes 🗌 1 | |
| | past 12 months (from date of | No 🗌 2 | SKIP to Q |
| | admission) | | |
| 33. | Number of changes in ART | One 1 | |
| | regimen in past 12 months | Two 2 | |
| | regimen in past 12 months | Three 3 | |
| FIR | ST change in ART regimen in the las | t 12 months from date of admission. Must be d | lifferent from CURRENT |
| | reg | gimen. Source: electronic database | |
| 34. | First two drugs ('NRTI backbone') | ABC/3TC 1 | |
| | listed in the CURRENT ART | AZT/3TC 2 | |
| | regimen: | TDF/3TC 3 | |
| | regimen. | Other, specify: 88 | |
| | | Unknown/not documented 🗌 87 | |
| 35. | Third drug listed in the CURRENT | NVP 1 | |
| | ART regimen: | EFV 2 | |
| | | ATV/r 🔲 3 | |
| | | LPV/r ☐ 4 | |
| | | DTG 5 | |
| | | DRV 🔲 6 | |
| | | Other, specify: 88 | |
| | | Unknown/not documented 87 | |
| 36. | ART regimen start date | Known 📙 1 | |
| | (dd/mm/yyyy) | Date: / / | |
| | | Unknown/not documented 🗌 87 | |
| 37. | ART regimen stop date | Known 1 | |
| | (dd/mm/yyyy) | Date: / / | |
| | | Unknown/not documented 🗌 87 | |
| 38. | Reason for stopping | Side effects 1 | |
| | | Treatment failure 🗌 2 | |
| | | Drug interactions (e.g., TB treatment) 3 | |
| | | Pregnancy 🗌 4 | |
| | | Change in treatment protocol 5 | |
| | | Other, specify: 88 | |
| | | Unknown/not documented 87 | |
| | <b>SECOND</b> change in ART Regimen in | the last 12 months from date of admission. Mu | ist be different from |
| | CURREN | IT regimen. Source: electronic database | |
| 39. | First two drugs ('NRTI backbone') | ABC/3TC 1 | |
| | listed in the CURRENT ART | AZT/3TC 2 | |
| | regimen: | TDF/3TC 3 | |
| | | Other, specify: 88 | |
| | | Unknown/not documented 🗌 87 | |
| 40. | Third drug listed in the CURRENT | NVP 1 | |
| | ART regimen: | EFV 🔲 2 | |
| | | ATV/r 🔲 3 | |
| | | LPV/r ∐ 4 | |
| | | DTG 📙 5 | |

| | | DRV 🔲 6 | |
|---|---|---|---|
| | | Other, specify: 88 | |
| | | Unknown/not documented 🗌 87 | |
| 41. | ART regimen start date | Known 1 | |
| | (dd/mm/yyyy) | Date: / / / | |
| | | Unknown/not documented 🗌 87 | |
| 42. | ART regimen stop date | Known 1 | |
| | (dd/mm/yyyy) | Date: / / / | |
| | | Unknown/not documented 🗌 87 | |
| 43. | Reason for stopping | Side effects 1 | |
| | | Treatment failure 2 | |
| | | Drug interactions (e.g., TB treatment) 3 | |
| | | Pregnancy 🗌 4 | |
| | | Change in treatment protocol 🗌 5 | |
| | | Other, specify: 88 | |
| | | Unknown/not documented 🗌 87 | |
| THI | | st 12 months from date of admission. Must be | different from CURRENT |
| | reg | gimen. Source: electronic database | |
| 44. | First two drugs ('NRTI backbone') | ABC/3TC 1 | |
| | listed in the CURRENT ART | AZT/3TC 2 | |
| | regimen: | TDF/3TC \[ 3 | |
| | | Other, specify: 88 Unknown/not documented 87 | |
| 45. | Third drug listed in the CURRENT | NVP 1 | |
| 45. | ART regimen: | EFV 2 | |
| | ANT Tegimen. | ATV/r 3 | |
| | | LPV/r 🗍 4 | |
| | | DTG 5 | |
| | | DRV` ☐ 6 | |
| | | Other, specify: 88 | |
| | | Unknown/not documented 87 | |
| 46. | ART regimen start date | Known 📙 1 | |
| | (dd/mm/yyyy) | Date:// | |
| 47 | ADT : | Unknown/not documented 87 | |
| 47. | ART regimen stop date | Known 📙 1 | |
| | (dd/mm/yyyy) | Date:// | |
| 40 | December to story in a | Unknown/not documented 87 | |
| 48. | Reason for stopping | Side effects 1 Treatment failure 2 | |
| | | Drug interactions (e.g., TB treatment) 3 | |
| | | Pregnancy 4 | |
| | | l | |
| | | Change in treatment protocol 5 | |
| | | Other, specify: 88 Unknown/not documented 87 | |
| | Pro-eynosure I | Prophylaxis (PrEP), Source: electronic database | |
| 49. | | Yes 1 | |
| +3. | Receipt of PrEP in pregnancy (indicated from log) | No 2 | END |
| | imalcatea ji oili logj | Unknown/not documented 87 | LIND |
| 50. | PrEP regimen | TDF + 3TC 1 | |
| , JJ. | | 101 1310 🔲 1 | 1 |

| | | Cabotegravir (injection) 2 | |
|---|---|---|---|
| | | Dapivirine 3 | |
| | | Unknown/not documented 🗌 87 | |
| 51. | Date started PrEP | Known 1 | |
| | (dd/mm/yyyy) | Date:// | |
| | | Unknown/not documented 🗌 87 | |
| 52. | Date stopped PrEP | Known 1 | |
| | (dd/mm/yyyy) | Date:/ / | |
| | | Unknown/not documented 🗌 87 | |
| 53. | Select yes if abortion | Yes 1 | |
| | | No 🗌 2 | Select 'Yes' if it's an |
| | | | abortion and the |
| | | | woman is available for |
| | | | an interview. If yes, |
| | | | conduct entire |
| | | | interview. |
| | | | Select "No" if it is an |
| | | | abortion and women is |
| | | | not available for an |
| | | | interview. If "No", skip |
| | | | to PART V: BIRTH |
| | | | DEFECT QUESTIONS on |
| | | | the women interview |
| | | | form. |

| Eswatini Birth Outcomes Study | Participant Number: | |
|---|---|---|
| Assessment of Birth Outcomes in Fountini for | .llavvina Transition to | Dalutarus in based Treatment |

## Assessment of Birth Outcomes in Eswatini following Transition to Dolutegravir-based Treatment Women Interview Form for Suspected Birth Defects

| MATERNITY NAME | |
|---|---|
| | Mbabane Government Hospital 🔲 1 |
| Raleigh Fitkin Memorial Hospital | |
| GOOD SHEPHERD HOSPITAL | |
| HLATIKHULU HOSPITAL | |
| | Mankayane Government Hospital 5 |
| INTERVIEWER'S NAME/ID: | DAY / MONTH / YEAR OF INTERVIEW: |
| NAME: | //2_0 |
| ID: | |
| INDICATE IF; | LIVE/STILLBIRTH, START FROM PART 1 |
| | MEDICAL ABORTION, WOMEN AVAILABLE, START FROM PART 1 |
| | MEDICAL ABORTION, WOMEN NOT AVAILABLE GO TO PART V: |

## PART I. MATERNAL CHARACTERISTICS AND HEALTH HISTORY

| Instructions: I will start with questions about your pregnancy history. I will ask you questions but also verify in your records as we go along. | | | | |
|---|---|---|---|--|
| 1.1 | Nationality | Eswatini 1 1 Other, specify: 88 | | |
| 1.2 | Date of last menstrual period (dd/mm/yyyy) | From records:/ 1 Estimated:/ 2 | | |
| 1.3 | Gestational age at booking | weeks, days 1 Don't know/not documented 87 | | |
| 1.4 | Mother's weight at first ANC | Kgs | | |
| 1.5 | Mother's most recent weight | At last ANC Kgs | | |
| 1.6 | Mother's height at ANC | Cm | | |
| 1.7 | Gravida | # of pregnancies | _ | |
| 1.8 | Parity | # of births ☐ 1<br>Don't know ☐ 87 | |
|---|---|---|---|
| 1.9 | Have you had any previous preterm deliveries (about < 37 weeks gestation)? | Yes | |
| 1.10 | Have you had any previous stillborn children? | Yes ☐ 1<br>No ☐ 2<br>Don't know ☐ 87<br>N/A ☐ 99 | |
| 1.11 | How many birth defects have you had in your previous pregnancies? | None | |
| 1.12 | If yes, please specify birth defect(s) or describe (if name unknown) | | |
| HIV-REL/ | ATED HISTORY | | |
| 1.13 | When was your most recent HIV test done? | Before pregnancy 1 During pregnancy, before delivery 2 At labor and delivery 3 After delivery, before hospital discharge 4 Don't know 87 | |
| 1.14 | What is your HIV status? | HIV positive 1 HIV negative 2 Don't know 87 Never tested for HIV 4 | SкIP ТО Q<br>SкIP ТО Q<br>SкIP ТО Q |
| 1.15 | When was your first positive HIV test? | /(dd/mm/yyyy) | |
| 1.16 | When was your most recent HIV negative test? | /(dd/mm/yyyy) | |
| 1.17 | When did you initiate ART? | / (dd/mm/yyyy) | |
| DΔRT | II. HIV-RFLATED DRUG USF | | |

Instructions (to say to participant): For this and subsequent questions, we are interested in learning more about what health conditions you have and what medicines you took before and after pregnancy. I will start with asking about HIV medicines, for treatment or prophylaxis. Then, I will ask about any medical conditions and other medicines, selected behaviors and any pregnancy complications. Finally, I will talk to you about the baby and birth and information on the suspected birth defect.

| <b>For interviewers,</b> please note: <u>Before pregnancy</u> refers to the time from the month before pregnancy based on LMP or best estimate. This section should be skipped for HIV negative women. | | | |
|---|---|---|---|
| 2.1 | Is there documentation of ANY ARVs initiated or continued during this pregnancy? | Yes 1<br>No 2 | Sкір то Q |
| 2.2 | Is there documentation of ARVs at the time of conception? | Yes, ART | If '2' Skip to<br>Q2.32 |
| 2.3 | Initial regimen prescribed or continued during pregnancy | TDF+3TC | |
| 2.4 | Start date of initial regimen: dd/mm/yyyy | // | |
| 2.5 | Indicate if any part of the date is estimated (can select more than one if a 'Yes' response is selected) | No 1<br>Yes, day 2<br>Yes, month 3<br>Yes, year 4 | |
| 2.6 | Is there documentation of change of ARVs to a new regimen during pregnancy? | Yes 1<br>No 2 | SKIP ТО Q |
| 2.7 | How many times were ARVs changed during pregnancy? | One | |
| 2.8 | Date of first change of ARV regimen: dd/mm/yyyy | // | |
| 2.9 | Indicate if any part of the date is estimated (can select more than one if a 'Yes' response is selected). | No 1<br>Yes, day 2<br>Yes, month 3<br>Yes, year 4 | |
| 2.10 | Reason for first change of ARV regimen? | Side effects 1 Treatment failure 2 Drug interactions (e.g., TB treatment) 3 Pregnancy 4 Change in treatment protocol 5 Other, specify: 88 Don't know/not documented 87 | |
| 2.11 | Second ARV regimen in pregnancy? | TDF+3TC+EFV | |

| 2.12 | Date of second change of ARV regimen: dd/mm/yyyy | // |
|---|---|---|
| 2.13 | Indicate if any part of the date is estimated (can select more than one if a 'Yes' response is selected) | No |
| 2.14 | Reason for second change of ARV regimen? | Side effects 1 Treatment failure 2 Drug interactions (e.g., TB treatment) 3 Pregnancy 4 Change in treatment protocol 5 Other, specify: 88 Don't know/not documented 87 |
| 2.15 | Third ARV regimen in pregnancy? | TDF+3TC+EFV |
| 2.16 | Date of third change of ARV regimen: dd/mm/yyyy | // |
| 2.17 | Indicate if any part of the date is estimated (can select more than one if a 'Yes' response is selected) | No |
| 2.18 | Reason for third change of ARV regimen? | Side effects 1 Treatment failure 2 Drug interactions (e.g., TB treatment) 3 Pregnancy 4 Change in treatment protocol 5 Other, specify: 88 Don't know/not documented 87 |
| 2.19 | Fourth ARV regimen in pregnancy? | TDF+3TC+EFV 1<br>TDF+3TC+DTG 2<br>AZT+3TC+DTG 3<br>AZT+3TC+EFV 4<br>Other, specify: 88 |
| 2.20 | Date of fourth change of ARV regimen: dd/mm/yyyy | // |
| 2.21 | Indicate if any part of the date is estimated (can select more than one if a 'Yes' response is selected) | No |
| 2.22 | During the time of your last menstrual period, did you miss any days taking your ARVS? | Yes |

| 2.23 | Is there documentation of termination or defaulting of ARVs during pregnancy? (stopping ARVs and not starting onto a new regimen prior to delivery) Yes responses include women not on ARVs at time of delivery but previously on ARVs in pregnancy | Yes | ЅкіР ТО Q |
|---|---|---|---|
| 2.24 | Date of ARV termination/defaulting date: dd/mm/yyyy | // | |
| 2.25 | Indicate if any part of the date is estimated (can select more than one if a 'Yes' response is selected). | No | |
| 2.26 | Comments (please provide any ARV related clarifications or explanations for a disruption of ARVs >1 week). | | |
| 2.27 | Did you take any other medicine (including traditional medicine) or therapy? | Yes 🔲 1<br>No 🔲 2 | Sкір то Q |
| 2.28 | If yes, first medicine/therapy: | | |
| 2.29 | First medicine/therapy: When did you take it? (multiple responses permitted in some cases) | Up to a month before pregnancy 1 In 1 <sup>st</sup> trimester 2 In 2 <sup>nd</sup> trimester 3 In 3 <sup>rd</sup> trimester 4 Don't know if before or during pregnancy 5 During pregnancy, but don't know trimester 6 | |
| 2.30 | If yes, second medicine/therapy: | No second therapy 99 | SKIP TO Q |
| 2.31 | Second medicine/therapy: When did you take it? (multiple responses permitted in some cases) | Up to a month before pregnancy 1 In 1st trimester 2 In 2nd trimester 3 In 3rd trimester 4 Don't know if before or during pregnancy 5 During pregnancy, but don't know trimester 6 | |

| 2.32 | If on PrEP, PrEP regimen | | | | | TDF+3T<br>ravir (injection<br>Dapivirin<br>ot documente | a) | |
|---|---|---|---|---|---|---|---|---|
| 2.34 | Date started PrEP (dd/mm/yyyy) | | | Known 1 Date: / / 87 | | | | |
| 2.35 | Date stopped PrEP (dd/mm/yyyy) | | | | | Know<br>_ / /<br>ot documente | | |
| DAD | T III. RISK FACTORS | | | | | | | |
| | NUTRIENTS | | | | | | | |
| | Micronutrient Use | No | Yes, but unknow | wn timing | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
| 3.1 | FOLIC ACID | | Don't know i<br>during pregr<br>During preg<br>don't know trim | nancy 🔲 1<br>nancy, but | | | | |
| 3.2 | Multivitamin | | during pregr | Don't know if before or during pregnancy 1 During pregnancy, but | | | | |
| 3.3 | Ferrous Sulfate<br>(Iron) | | Don't know i<br>during pregr<br>During preg<br>don't know trim | nancy 🔲 1<br>nancy, but | | | | |
| DIABET | ·FS | | | | | | | |
| 3.4 | Do you currently have | e diabete | rs? | | | Don | Yes ☐ 1<br>No ☐ 2<br>'t know ☐ 87 | |
| 3.5 | Did you have diabete | Yes ☐ 1<br>No ☐ 2<br>Don't know ☐ 87 | | | | | | |
| 3.6 | .6 If yes to 3.4, what medicines for your diabetes did you take very early in this pregnancy between your first and third month of pregnancy? (Response should exclude traditional medicines) | | | None | | | | |
| 3.7 | If yes to 3.4, were you in control during this | | | | Yes | | | |

**CONVULSIONS (EPILEPSY)** 3.8 Have you ever had convulsions? Yes 1 SKIP TO Q No  $\square$  2 SKIP TO Q ገ 87 Don't know 3.9 Did you have convulsions just before you got pregnant? Yes 1 No 2 Don't know 87 Yes 1 3.10 Did you have any convulsions during this pregnancy? No □ 2 Don't know ☐ 87 Yes, 1st Yes, 2<sup>nd</sup> Yes, 3rd Medicines used for Yes, but unknown timing Yes, Before No pregnancy trimester trimester trimester convulsions (Epilepsy) 3.11 VALPROIC ACID Don't know if before or (DEPAKENE) during pregnancy 1 During pregnancy, but don't know trimester 2 PHENYTOIN (DILANTIN) 3.12 Don't know if before or during pregnancy 1 П During pregnancy, but don't know trimester 2 Don't know if before or 3.13 FELBAMATE (FELBATOL) during pregnancy 1 During pregnancy, but don't know trimester 2 3.14 **C**ARBAMAZEPINE Don't know if before or (TEGRETOL) during pregnancy 1 П During pregnancy, but don't know trimester 2 Don't know if before or 3.15 **PHENOBARBITAL** during pregnancy | 1 (LUMINAL) П During pregnancy, but don't know trimester 2 3.16 OTHER MEDICINE, Don't know if before or SPECIFY: during pregnancy 1 During pregnancy, but don't know trimester 2 **MALARIA** Did you have malaria during this pregnancy? Yes 1 3.17 SKIP TO Q No **□** 2 SKIP TO Q Don't know ∃ 87 3.18 Did you take any medicines or remedies for Yes 1 malaria during this pregnancy? SKIP TO Q No 2 SKIP TO Q Don't know 87

| | Medicines used for<br>Malaria | No | Yes, but unknow | n timing | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
|---|---|---|---|---|---|---|---|---|
| 3.19 | Coartem<br>(artemether/<br>LUMAFANTRINE) | | Don't know if b<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy <u>,</u> but | | | | |
| 3.20 | Duocotexin<br>(dihydroartemisinin/<br>piperaquine) | | Don't know if b<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy, but | | | | |
| 3.21 | Fansidar | | Don't know if k<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy, but | | | | |
| 3.22 | Quinine | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.23 | UNKNOWN MEDICINE | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.24 | OTHER MEDICINE, SPECIFY: | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| TURFRC | CULOSIS | | | | | | | |
| 3.25 | Did you have tuberculd pregnancy? | osis duri | ng this | | Dor | Yes 1<br>No 2<br>n't know 8 | SKIP TO Q SKIP TO Q | |
| 3.26 | Did you take any medic<br>tuberculosis during this | | | | Dor | Yes | SKIP TO Q<br>SKIP TO Q | |
| | Medicines used for TB | No | Yes, but unknow | n timing | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
| 3.27 | INH | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.28 | Rifampin | | Don't know if k<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy, but | | | | |

| | Medicines used for TB | No | Yes, but unknown | n timing | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
|---|---|---|---|---|---|---|---|---|
| 3.29 | Pyrazinamide (PZA) | | Don't know if k<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy, but | | | | |
| 3.30 | ETHAMBUTOL | | Don't know if k<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy <u>, b</u> ut | | | | |
| 3.31 | Streptomycin | | Don't know if t<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy, but | | | | |
| 3.32 | Unknown medicine | | Don't know if t<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy, but | | | | |
| 3.33 | OTHER MEDICINE, SPECIFY: | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| FEVER | | | | | | | | |
| 3.34 | | | | Yes ☐ 1<br>No ☐ 2<br>Don't know ☐ 87 | | | | |
| 3.35 | Did you have fevers are pregnant? | | | | Dor | Yes 🗌 1<br>No 🔲 2<br>n't know 🔲 8 | SKIP TO Q<br>SKIP TO Q | |
| 3.36 | Did you take any medic<br>fever? | cines or | remedies for the | | Dor | Yes 1<br>No 2<br>n't know 8 | SKIP TO Q<br>SKIP TO Q | |
| | Medicines used for<br>Fever | No | Yes, but unknown | n timing | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
| 3.37 | Aspirin | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.38 | Paracetamol<br>(Panadol) | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.39 | Ibuprofen (Brufen) | | Don't know if t<br>during pregna<br>During pregna<br>don't know trimes | ncy 🔲 1<br>ancy <u>, b</u> ut | | | | |

| | Medicines used for<br>Fever | No | Yes, but unknown timin | ng | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
|---|---|---|---|---|---|---|---|---|
| 3.40 | Diclofenac | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.41 | OTHER MEDICINE, SPECIFY: | | Don't know if before during pregnancy During pregnancy, b | ] 1 | | | | |
| ANTIBIC<br>3.42 | DTIC USE Did you take antibio | tics for | anything other than | | | | Yes 1 | |
| 3.42 | fever during this pre | | - | | | Don' | No 2 2 | SKIP TO Q<br>SKIP TO Q |
| 3.43 | If yes, for what cond | lition? | | | Specify: | | 1 | |
| | | | | | | | t know 🗌 87 | |
| | Antibiotics | No | Yes, but unknown timir | ng | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
| 3.44 | Ciprofloixacin | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.45 | CEFTRIAXONE | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.46 | ERYTHROMYCIN | | Don't know if before during pregnancy During pregnancy, but doknow trimester | ] 1 | | | | |
| 3.47 | Amoxicillin | | Don't know if before<br>during pregnancy<br>During pregnancy, but do<br>know trimester | ] 1<br>on't | | | | |
| 3.48 | Doxycycline | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.49 | Penicillin | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| 3.50 | CLOXACILLIN | | Don't know if before during pregnancy During pregnancy, but do | ] 1<br>on't | | | | |

| | Antibiotics | No | Yes, but unknow | wn timing | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
|---|---|---|---|---|---|---|---|---|
| 3.51 | Fluconazole | | Don't know<br>during preg<br>During pregnancy<br>know trim | nancy 🔲 1<br>y, but don't | | | | |
| 3.52 | COTRIMOXAZOLE | | Don't know<br>during preg<br>During pregnancy<br>know trim | nancy 🔲 1<br>y, but d <u>on</u> 't | | | | |
| 3.53 | OTHER, SPECIFY: | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| ANY OT | HER DRUG/THERAPY US | SE | | | | | | |
| | Please use the space be from the month before | elow to | • | _ | - | | fore pregnancy | (= time |
| | Other | No | Yes, but unknow | | Yes, Before pregnancy | Yes, 1 <sup>st</sup><br>trimester | Yes, 2 <sup>nd</sup><br>trimester | Yes, 3 <sup>rd</sup><br>trimester |
| 3.54 | | | Don't know if<br>during pregn<br>During pregr<br>don't know trime | ancy 🔲 1<br>nancy, but | | | | |
| 3.55 | | | Don't know if before or during pregnancy 1 During pregnancy, but don't know trimester 2 | | | | | |
| TRADIT | IONAL MEDICINE | | | | | | | |
| 3.56 | Did you take any trac<br>before pregnancy or<br>pregnancy? | | _ | | | Dor | Yes | SKIP TO Q<br>SKIP TO Q |
| 3.57 | Select all that apply. | what condition did you take it for? Ill that apply. The next two questions asked for each condition indicated | | | Diabetes 1 | | | |
| 3.58 | Indicate the name or medicine. | main in | gredient of the | Specify: | | | | |
| 3.59 | When did you take it | ? | | During ( | | During first to<br>uring second to<br>During third to<br>Before pro | rimester 2 2 rimester 3 egnancy 4 | May have<br>multiple<br>responses<br>to 1-5; if<br>select 6, |

| | | Don't know if before or during pregnancy | 6 should be only response |
|---|---|---|---|
| BEHAVI | ORAL RISK FACTORS | | |
| 3.60 | How often did you consume alcohol during pregnancy? | Never Occasionally Sometimes Frequently | 1<br>2<br>3<br>4 |
| 3.61 | How often did you smoke cigarettes or use other tobacco products during pregnancy? | Never Occasionally Sometimes Frequently | 1<br>2<br>3<br>4 |
| PREGNA | ANCY COMPLICATIONS AND COVID-19 | | |
| 3.62 | Maternal diagnoses/complications during pregnancy (select all that apply) | None 1 Pre-eclampsia 2 Hypertension 3 Diabetes mellitus 4 Excess weight gain, obesity 5 Syphilis 6 High blood pressure 7 Other, specify: | |
| 3.63 | Hemoglobin at ANC | Hgb at first ANC: 1 Hgb at other ANC visit (if 1 <sup>st</sup> not available): 2 Don't know 87 | |
| 3.64 | Were you diagnosed with COVID-19 during this pregnancy? | Yes | KIP TO Q |
| 3.65 | If yes, how was it diagnosed? | COVID-19 test done 1 Diagnosis based on symptoms only 2 Other, specify: 88 | |
| 3.66 | If yes, what trimester were you diagnosed? | First 1 Second 2 Third 3 Don't know 87 | |
| PART | IV. INFANT AND DELIVERY OUTCOME | S | |
| | Instructions: I will now ask you questions all questions while also verifying in your reco | bout the birth (and child if NOT still born). As before, I words. | vill ask you |
| 4.1 | Gestational age at delivery (or at time of medical induced abortion) | weeks, days 1 Don't know/not documented 87 | |

| 4.2 | Single or multiple birth | Single 1 Twin 2 | Qs should repeat<br>for second and<br>third births |
|---|---|---|---|
| | | Triplet 3 | tillia birtiis |
| 4.3 | Date of birth or abortion (dd/mm/yyyy) | // | |
| 4.4 | Type of birth | Liveborn 1 Stillborn 2 Medically Induced Abortion 3 | |
| 4.5 | Birth weight | grams 1<br>Don't know 87 | |
| 4.6 | Child sex | Male 1<br>Female 2<br>Ambiguous 3 | For abortion and stillbirth, Q should be answered, then skip to Q4.11 |
| 4.7 | Length | cm 1<br>Don't know 87 | |
| 4.8 | Head circumference | cm 1<br>Don't know 87 | |
| 4.9 | Apgar score | | |
| 4.10 | Newborn complications | Jaundice 1 Hypoglycemia 2 Resuscitation 3 Other, specify: 88 | |
| 4.11 | Date birth defect identified (dd/mm/yyyy) | // | |
| PART | V. BIRTH DEFECT QUESTIONS | | |
| 5.1 | One or more abnormalities identified: | First infant born | Skip pattern to go<br>to the affected<br>child(ren) |
| 5.2 | Is the abnormality an extra digit? | Yes | SKIP TO Q |
| 5.3 | Where are the extra digits? (select all that apply) | Left hand 1 Right hand 2 Left foot 3 Right foot 4 Don't know 87 | |

| 5.4 | Where on the left hand is the extra digit located? | Near the fifth digit (pinky finger) 1 Near the thumb 2 Other place, specify: 88 | |
|---|---|---|---|
| 5.5 | Does the extra digit appear as: | A fullly formed extra digit (seems to look like a finger and have bone in it) 1 Soft, without a bone (sometimes hanging by a stalk) 2 | |
| 5.6 | Where on the right hand is the extra digit located? | Near the fifth digit (pinky finger) | |
| 5.7 | Does the extra digit appear as: | A fullly formed extra digit (seems to look like a finger and have bone in it) 1 Soft, without a bone (sometimes hanging by a stalk) 2 | |
| 5.8 | Where on the left foot is the extra digit located? | Near the fifth digit (pinky toe) 1 Near the big toe 2 Other place, specify: 88 | |
| 5.9 | Does the extra digit appear as: | A fullly formed extra digit (seems to look like a finger and have bone in it) 1 Soft, without a bone (sometimes hanging by a stalk) 2 | |
| 5.10 | Where on the right foot is the extra digit located? | Near the fifth digit (pinky toe) 1 Near the big toe 2 Other place, specify: 88 | |
| 5.11 | Does the extra digit appear as: | A fullly formed extra digit (seems to look like a finger and have bone in it) 1 Soft, without a bone (sometimes hanging by a stalk) 2 | |
| 5.12 | Please provide any other details on this abnormality that are not captured above. | Description: | |
| 5.13 | Is the head and neck exam NORMAL? (includes skull, fontanelles, eyes, ears, nose, jaw) | Yes 1<br>No 2<br>Don't know 87 | SKIP TO Q |

| 5.14 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
|---|---|---|---|
| 5.15 | Is there evidence of hydrocephalus (swollen head)? | Yes 1<br>No 2<br>Don't know 87 | |
| 5.16 | Is there a defect in the skull? | Yes | |
| 5.17 | If there is a defect in the skull, is it: | Completely covered by skin 1 Partly covered by skin 2 Covered by a thin sac/membrane 3 Not covered by skin (brain tissue visible) 4 Don't know 87 | |
| 5.18 | Is the mouth, lip and palate exam NORMAL? (cleft lip or palate) | Yes 1<br>No 2<br>Don't know 87 | SKIP ТО Q |
| 5.19 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
| 5.20 | Is the chest exam NORMAL? (shape and respiratory movements) | Yes 1<br>No 2<br>Don't know 87 | SKIP TO Q |
| 5.21 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
| 5.22 | Are the abdominal and anal exam NORMAL? (masses/anal closure defect) | Yes | SKIP TO Q |

| 5.23 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
|---|---|---|---|
| 5.24 | Are the arms and legs NORMAL? (length, shape, missing parts) | Yes | SKIP TO Q |
| 5.25 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
| 5.26 | Are the fingers and toes NORMAL? (including nails, number, dangling fused, shape or parts missing, abnormally large or small) | Yes | SKIP TO Q |
| 5.27 | If no, please describe abnormality: (please include as much detail as possible) | Description: | |
| | If not known, explain why: | | |
| 5.28 | Is the Spine exam NORMAL? (lumps or cysts or bulging in the back including the neck, thorax or lumbar area) | Yes | Sкір То Q |
| 5.29 | If no, please describe abnormality: (please include as much detail as possible) If unknown, explain why: | Description: | |

| 5.30 | Where in the spine is the defect located? (Select all that apply) | Cervical 1<br>Thoracic 2<br>Lumbosacral 3<br>Don't know 87 | |
|---|---|---|---|
| 5.31 | Is the spinal defect: | Covered in hair and NOT bulging out 1 Covered in hair and bulging out 2 Bulging out and completely covered with skin 3 Bulging out and partly covered with skin 4 Bulging out and covered with only a sac/thin membrane 5 Open-can see the spine/spinal cord 6 Don't know 87 | |
| 5.32 | Are the hips and genitalia NORMAL? (including urethra, testes, penile shaft, vagina, labia) | Yes | SKIP TO Q |
| 5.33 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
| 5.34 | Is the skin exam NORMAL? (pale, blue, birth marks, or any large very red areas) | Yes | SKIP TO Q |
| 5.35 | If no, please describe abnormality: (please include as much detail as possible) If not known, explain why: | Description: | |
| 5.36 | Describe any other abnormality, unusual finding or make any comment about abnormality | Description: | |

| 5.37 | Please indicate the preliminary diagnosis for this child. | Central nervous system: Anencephaly |
|---|---|---|
| | | Eye and ear malformations: Anophthalmia 8 Microphthalmia 9 Anotia 10 |
| | | Microtia 11 Orofacial clefts: Cleft lip 12 Cleft palate 13 Cleft lip and palate 14 |
| | | Malformations of digestive system and genital organs Imperforate anus 15 Hypospadias 16 |
| | | Musculoskeletal: Talipes equinovarus / Clubfoot |
| | | Gastroschisis |
| 5.38 | Confirm that a doctor has reviewed and approved of the responses in section 5. | Yes |
| 5.39 | Providers completing or providing input on this form (list all that apply) | Doctor name:<br>Midwife name:<br>Other: |

| Α | В | С | D | E | F- | G | H | | J | K | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| watini Birth | Outcomes Stu | ıdy | | | | | | | | | |
| rth Defects S | pecialist Eval | uation Form, Version 2.0, 17 Novembe | er 2021 | | | | | | | | |
| ate Sent | PTID | Preliminary (Interview) diagnosis | If other, specify | Interview Description (optional) | Instance (photo file) if available | Reviewer Defect Description | Organ system | If other, specify | Organ System/Preferred Term | Final defect determination | Comments |
| | | ,, , , | | , | , | | . , | | 0 , . | | |